A Phase 1, Single-Center, Randomized, 3-Period Crossover Study in Healthy Volunteers to Evaluate the Absorption of WTX101 After Single Dose Administration of an Enteric Coated Formulation with and without food and a Non-Coated Formulation Coadministered with a Proton Pump Inhibitor without Food

**Unique Protocol ID:** WTX101-102

NCT Number: NCT05319912

**Date of SAP:** 22 May 2014



- 16.1.9 **Documentation of Statistical Methods**
- 16.1.9.1 Pharmacokinetic Analysis
- 16.1.9.1.1 Pharmacokinetic Analysis Plan

# A Phase 1, Single-Center, Randomized, 3-Period Crossover Study in Healthy Volunteers to Evaluate the Absorption of WTX101 After Single Dose Administration of an Enteric Coated Formulation with and without food and a Non-Coated Formulation Coadministered with a Proton Pump Inhibitor without Food

# Protocol WTX101-102

# Pharmacokinetic Analysis Plan

Version 1 May 22, 2014

Prepared for: WilsonTherapeutics USA, Inc.

P.O. Box 17757

Urbana, Illinois 61803

USA

Wilson Therapeutics, AB Västra Trädgårdsgatan 15

11453 Stockhold

Sweden

Prepared by: Kramer Consulting LLC

14313 Outpost Way

North Potomac, MD 20878

## SIGNATURE PAGE



WilsonTherapeutics USA, Inc.

# Table of Contents

| | | Page |
|---|---|---|
| | Signature Page | i |
| | Table of Contents | . ii |
| | List of Abbreviations | iii |
| 1.0 | Introduction | . 1 |
| 2.0 | Study Overview | . 1 |
| 3.0 | Pharmacokinetic Sampling Schedule | . 2 |
| 4.0 | Blinding and Unblinding. | . 3 |
| 5.0 | Interim Analysis | . 3 |
| 6.0 | Pharmacokinetic Analysis | . 3 |
| 6.1<br>6.2<br>6.2.1 | Analysis Population | . 3 |
| 7.0 | Statistical Analyses | . 4 |
| 7.1<br>7.2<br>7.3 | Primary Analysis Secondary Analysis Exploratory Analysis | . 5 |
| 8.0 | Quality Control Procedures | . 6 |
| 9.0 | Tables, Figures, Appendices | . 6 |
| 9.1<br>9.2<br>9.3 | Tables | . 6 |

#### List of Abbreviations

<u>Term</u> <u>Definition</u>

ANOVA Analysis of Variance

AUC(0-t) Area under the plasma concentration-time curve from 0 to the final

time with a concentration  $\geq$  LOQ

AUC(inf) Area under the plasma concentration-time curve from 0 to infinity

BMI Body Mass Index CI Confidence interval

CL/F Clearance uncorrected for bioavailability

Cmax Maximum plasma concentration

EC Enteric coated F Bioavailability

GMR Geometric mean ratio

h Hour

IM Intramuscular kg Kilogram

LOQ Validated lower limit of the bioanalytical method

m² Squared meter
mg Milligram
mL Milliliter
Mo Molybdenum
MSE Mean squared error

ng Nanogram

PK Pharmacokinetic

PKAP Pharmacokinetic analysis plan

PPI Proton pump inhibitor SAP Statistical analysis plan t½ Elimination half-life

Tmax Time of maximum plasma concentration

Vz/F Volume of distribution uncorrected for bioavailability

WSCV Within-subject coefficient of variation

λz Elimination rate constant

#### 1.0 Introduction

This pharmacokinetic analysis plan (PKAP) summarizes the planned presentation and analysis of the clinical pharmacokinetic data from WilsonTherapeutics USA, Inc. Protocol WTX101-102, "A Phase 1, Single-Center, Randomized, 3-Period Crossover Study in Healthy Volunteers to Evaluate the Absorption of WTX101 After Single Dose Administration of an Enteric Coated Formulation with and without food and a Non-Coated Formulation Coadministered with a Proton Pump Inhibitor without Food".

Some of the analyses detailed here may be more detailed or in some aspects slightly different than those described in the protocol. In case of differences, this PKAP would supersede the pharmacokinetic sections in the protocol.

Only the pharmacokinetic analyses are described in this PKAP. The summaries of demographics, baseline characteristics, and safety are detailed in a separate statistical analysis plan (SAP) for this study.

# 2.0 Study Overview

This is an open-label, 3-treatment, 3-period, 6-sequence, single-dose, randomized crossover study of the pharmacokinetics and comparative bioavailability of WTX101 after administration of an enteric coated (EC) tablet versus an uncoated capsule with a proton pump inhibitor (PPI) and after administration of the EC tablet under fed and fasted conditions.

The treatments to be administered are as follows:

Treatment A: WTX101 EC tablets,  $60 \text{ mg} (2 \times 30 \text{mg})$  on Day 1 after an overnight fast.

Treatment B: WTX101 EC tablets, 60 mg (2 × 30mg) on Day 1, 30 minutes after the start of a high calorie / high fat breakfast, preceded by an overnight fast.

Treatment C: Omeprazole 20 mg (1 × 20 mg delayed-release capsule) once-daily (QD) on the mornings of Days -5 to -1 after an overnight fast, omeprazole 20 mg delayed-release capsule at Hour -1 on Day 1 after an overnight fast, and WTX101 uncoated capsules, 60 mg (2 × 30mg) at Hour 0 on Day 1.

Eighteen (18) healthy adult male and female volunteers will be randomly assigned to 1 of 6 treatment sequences, as shown in Table 1.

Table 1: Treatment Sequences.

| | Treatment* | | |
|----------|----------------------------|---|---|
| Sequence | Period 1 Period 2 Period 3 | | |
| 1 | A | В | C |
| 2 | В | C | A |
| 3 | C | A | В |
| 4 | В | A | C |
| 5 | A | C | В |
| 6 | C | В | A |

<sup>\*</sup>A = WTX101 EC tablets, 60 mg (2  $\times$  30mg) on Day 1 after an overnight fast; B = WTX101 EC tablets, 60 mg (2  $\times$  30mg) on Day 1, 30 minutes after the start of a high calorie / high fat breakfast, preceded by an overnight fast; C = Omeprazole 20 mg (1  $\times$  20 mg delayed-release capsule) once-daily (QD) on the mornings of Days -5 to -1 after an overnight fast, omeprazole 20 mg delayed-release capsule at Hour -1 on Day 1 after an overnight fast, and WTX101 uncoated capsules, 60 mg (2  $\times$  30mg) at Hour 0 on Day 1.

Serial blood samples for the measurement of the plasma concentrations of total molybdenum (Mo) will be obtained over a 192-hour period after each dose. There will be a minimum 14-day washout between the dosing in each period.

# 3.0 Pharmacokinetic Sampling Schedule

On Study Days 1, 15, and 29 (Periods 1, 2, and 3, respectively), blood samples for the determination of total Mo concentrations will be collected before and at 1, 2, 3, 3.5, 4, 4.5, 5, 6, 7, 7.5, 8, 8.5, 9, 9.5, 10, 12, 14, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 192 hours after dosing. Samples collected through 48 hours will be on an inpatient basis and from 72 through 192 hours on an outpatient basis. There will be a minimum 14-day washout between the dosing in each period.

There will be a total of 84 blood samples for pharmacokinetics per subject, 28 per treatment.

# 4.0 Blinding and Unblinding

This is an objective study and blinding is not required.

# 5.0 Interim Analysis

No interim analysis will be conducted.

# 6.0 Pharmacokinetic Analysis

#### 6.1 Analysis Population

The analysis population will consist of all subjects who complete at least 2 periods of the study and have data sufficient for the determination of PK parameters. Any subjects that are excluded from the analysis will be listed along with the reason for the exclusion.

# 6.2 Pharmacokinetic Analysis

Actual blood sampling times will be used in all PK analyses. Per protocol times will be used to calculate mean plasma concentrations for tabular and graphical displays. All PK calculations and generation of individual subject plasma concentration vs. time graphs will be done using SAS® for Windows® Version 9.3 or higher under Windows XP Professional or higher. Graphs of mean plasma concentration will be prepared using SigmaPlot for Windows Version 12.5 or higher.

#### **6.2.1** Pharmacokinetic Parameters

Pharmacokinetic parameters for total Mo will be calculated using non-compartmental analysis. Only plasma concentrations equal to or greater than the validated lower limit (LOQ) of the assay will be used in the pharmacokinetic analysis. Plasma concentrations < LOQ will be taken as 0 for the calculation of the descriptive statistics for plasma concentrations at each sampling time. For the PK analysis, plasma concentrations < LOQ that occur from pre-dose to the first concentration  $\ge$  LOQ will be taken as 0 and those that occur thereafter will be taken as missing.

Cmax and Tmax will be taken directly from the data. The elimination rate constant,  $\lambda z$ , will be calculated as the negative of the slope of the terminal log-linear segment of the

plasma concentration-time curve. The slope will be determined from a plot of the natural log of the terminal plasma concentrations against time; at least 3 terminal plasma concentration time points, beginning with the final concentration  $\geq$  LOQ, will be selected for the determination of  $\lambda z$  and the regression will have a coefficient of determination ( $r^2$ )  $\geq$  0.9000. The range of data to be used for each subject and treatment will be determined by visual inspection of a semi-logarithmic plot of concentration vs. time. Elimination half-life ( $t^{1/2}$ ) will be calculated according to the following equation:

$$t^{1/2} = \frac{0.693}{\lambda z}.$$

Area under the curve to the final sample with a concentration  $\geq$  LOQ [AUC(0-t)] will be calculated using the linear trapezoidal method and extrapolated to infinity [AUC(inf)] using

$$AUC(\inf) = AUC(0-t) + \frac{C_{tf}}{\lambda z}$$

where  $C_{tf}$  is the final concentration  $\geq LOQ$ .

Clearance (CL/F) and volume of distribution (Vz/F), uncorrected for bioavailability (F), will be calculated according to

$$CL/F = \frac{Dose}{AUC(\inf)}$$
 and  $Vz/F = \frac{Dose}{AUC(\inf) \times \lambda z}$ ,

respectively.

## 7.0 Statistical Analyses

Individual subject plasma total Mo concentrations, blood sampling times, and PK parameters will be listed by treatment group. Plasma concentrations and PK parameters will be summarized by treatment group using descriptive statistics. Summaries for plasma concentrations will include number, arithmetic mean, standard error, and coefficient of variation, geometric mean and coefficient of variation, and minimum,

median and maximum. Summaries for PK parameters will include number, arithmetic mean, standard deviation, and coefficient of variation, geometric mean and coefficient of variation, and minimum, median, maximum.

## 7.1 Primary Analysis

The PK parameters for total Mo — Cmax, AUC(0-t), and AUC(inf) —will be compared among treatments using an Analysis of Variance (ANOVA) statistical model with sequence, treatment, and period as the fixed effects and subject within sequence as a random effect, using the natural logarithms of the data.

Confidence intervals (90%) will be constructed for the least squares geometric treatment ratios (GMR) — Treatment B (WTX101 EC Tablet + Food)-to-Treatment A (WTX101 EC Tablet Fasted) and Treatment A (WTX101 EC Tablet Fasted)-to-Treatment C (WTX101 Uncoated Capsule + PPI Fasted) — of all 3 parameters using the natural log-transformed data and the two one-sided t-tests procedure. The GMRs and associated 90% confidence limits (CI) will be exponentiated back to the original scale.

## 7.2 Secondary Analysis

The within-subject coefficient of variation (WSCV) of Cmax, AUC(0-t), and AUC(inf) will be estimated using

$$WSCV = 100\% \times \sqrt{e^{MSE} - 1}$$

where MSE is the mean squared error from the ANOVA.

## 7.3 Exploratory Analysis

Relationships between CL/F and Vz/F and body size — weight (kg) and BMI (kg/m² — will be examined graphically for each treatment. If suggested by the graphs, regression models may be fit to the data.

# **8.0 Quality Control Procedures**

All data — random code\*, plasma concentrations, dosing and sampling dates and times — will be received electronically, either as SAS datasets or Excel workbooks; no data, at any time, will be entered by hand. The creation of the analysis data sets will be quality controlled by a visual inspection of a graph of each subject's plasma concentration vs. time data to ensure that there are no errors.

The data used to construct summary figures and tables will be created by the SAS programs used to either create the analysis data sets or to perform the pharmacokinetic analyses. Data will be transferred electronically to Excel workbooks, e.g. there will be no data transcription, from which the figures and tables will then be constructed. Figures and tables will be hyperlinked to Appendix listings containing the source data.

As a final check, data from a minimum of two subjects will be selected, analyzed manually in an Excel workbook, and the results verified against those created by the SAS programs.

#### 9.0 Tables, Figures, Appendices

#### 9.1 Tables

Table 1: Summary of total Mo pharmacokinetic parameters after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC tablets to healthy volunteers under fasted and fed conditions and a single 60 mg (2 × 30 mg) dose of WTX101 uncoated capsules with a PPI under fasted conditions.

Table 2: Statistical analysis of total Mo pharmacokinetic parameters after administration of a single 60 mg ( $2 \times 30$  mg) dose of WTX101 EC tablets to healthy volunteers under fasted and fed conditions and a single 60 mg ( $2 \times 30$  mg) dose of WTX101 uncoated capsules with a PPI under fasted conditions.

# 9.2 Figures

Figure 1: Mean plasma concentrations of total Mo administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC tablets to healthy volunteers under fasted and fed conditions — linear axes (left panel) and semi-logarithmic (right panel).

-

<sup>\*</sup> If not created by Kramer Consulting LLC.

Figure 2: Mean plasma concentrations of total Mo administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC tablets and a single 60 mg (2 × 30 mg) dose of WTX101 uncoated capsules with a PPI to healthy volunteers under fasted conditions conditions — linear axes (left panel) and semi-logarithmic (right panel).

# 9.3 Appendices

Appendix I: Randomization Code

Appendix II: Individual Subject Plasma Total Mo Concentrations

Appendix III: Individual Subject Blood Sampling Times

Appendix IV: Mean ± Standard Deviation Plasma Total Mo Concentrations

(ng/mL)

Appendix V: Individual Subject Total Mo Pharmacokinetic Parameters

Appendix VI: Descriptive Statistics for Total Mo Pharmacokinetic Parameters

Appendix VII: Statistical Analysis of Total Mo Pharmacokinetic Parameters

Appendix VIII: Individual Subject Plasma Total Mo Concentration vs. Time

Graphs — Linear Axes

Appendix IX: Individual Subject Plasma Total Mo Concentration vs. Time

Graphs — Semi-Logarithmic Axes<sup>†</sup>

<sup>&</sup>lt;sup>†</sup> Graphs include line segments indicating the range of data used to estimate  $\lambda z$ .

# 16.1.9.1.2 Pharmacokinetic Report

# A Phase 1, Single-Center, Randomized, 3-Period Crossover Study in Healthy Volunteers to Evaluate the Absorption of WTX101 After Single Dose Administration of an Enteric Coated Formulation with and without food and a Non-Coated Formulation Coadministered with a Proton Pump Inhibitor without Food

# **Study WTX101-102**

# Pharmacokinetic and Statistical Report

| Prepared for: | Wilson Therapeutics USA, Inc.<br>P.O. Box 17757<br>Urbana, IL 61803<br>USA |
|---|---|
| | Wilson Therapeutics, AB<br>Västra Trädgårdsgatan 15<br>111 53 Stockholm<br>Sweden |
| Prepared by: | PPD |
| | Kramer Consulting LLC 14313 Outpost Way |
| | North Potomac, MD 20878-4352 |
| Signature: | υ |
| | PPD |
| Date: | July 14, 2014 |

# Table of Contents

| | | <u>I</u> | Page |
|---|---|---|---|
| | Table of Content | S | i |
| | List of Tables | | . ii |
| | List of Figures | | iii |
| | List of Abbrevia | tions | .iv |
| 1.0 | Synopsis of Pharmacokinetic Results | | |
| 2.0 | Introduction | | 2 |
| 3.0 | Objective | | 2 |
| 4.0 | Study Conduct. | | 3 |
| 4.1<br>4.2<br>4.3 | Bioanalytical | c and Statistical Analyses | 3 |
| 5.0 | Overview of the | Study Design | 3 |
| 6.0 | Pharmacokineti | c and Statistical Methods | 4 |
| 6.1<br>6.2<br>6.2.1<br>6.2.2<br>6.2.3 | Statistical Meth<br>Primary Analys<br>Secondary Anal | e Methods ods is ysis alysis | 6<br>6<br>7 |
| 7.0 | Results | | 7 |
| 7.1<br>7.2<br>7.3<br>7.3.1<br>7.3.2 | Pharmacokinetic<br>Pharmacokinetic<br>Results | Pre-Dose Concentration ≥ LOQc Analysis Populationcs | 8<br>8 |
| 8.0 | Conclusions | | 16 |
| 9.0 | References | | 17 |
| | Appendix I Appendix II Appendix III Appendix IV Appendix V Appendix VI Appendix VIII Appendix VIII Appendix IX | Random Code Subject Height, Weight, and BMI Individual Subject Plasma Concentrations Individual Subject Blood Sampling Times Descriptive Statistics for Plasma Concentrations Individual Subject Pharmacokinetic Parameters Descriptive Statistics for Pharmacokinetic Parameters Statistical Analysis of Pharmacokinetic Parameters Individual Subject Total Mo Plasma Concentration vs. Time Graphs — Linear Axes Individual Subject Total Mo Plasma Concentration vs. | 19<br>20<br>26<br>32<br>35<br>38<br>39 |
| | Appendix A | Time Graphs — Semi-Logarithmic Axes | 51 |

Wilson Therapeutics USA, Inc. Study WTX101-102

Page ii July 14, 2014

# List of Tables

| | | Page |
|---|---|---|
| Table 1: | Treatment Sequences. | 4 |
| Table 2: | Subjects with a pre-dose concentration ≥ LOQ. | 8 |
| Table 3: | Summary of total Mo PK parameters after administration of a single $60 \text{ mg} (2 \times 30 \text{ mg})$ dose of WTX101 EC Tablets under fasted and fed conditions and UC + PPI under fasted conditions. | 12 |
| Table 4: | Statistical analysis of total Mo PK parameters after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC Tablets under fasted and fed conditions and UC + PPI under fasted conditions | 13 |
| Table 5: | Summary of between-subject coefficients of variation of total Mo Cmax, AUC(0-t), and AUC(inf) after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC Tablets under fasted and fed conditions and UC + PPI under fasted conditions | 15 |

# List of Figures

| | | <u>Page</u> |
|---|---|---|
| Figure 1: | Mean $\pm$ standard error plasma concentrations of total Mo after administration of a single 60 mg (2 $\times$ 30 mg) dose of WTX101 EC Tablets under fasted and fed conditions and UC + PPI under fasted conditions — linear axes (left panel) and semi-logarithmic (right panel). | 11 |
| Figure 2: | Individual subject CL/F vs. body weight (left panel) and BMI (right panel) of total Mo after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC Tablets fasted to healthy volunteers | 14 |
| Figure 3: | Individual subject CL/F vs. body weight (left panel) and BMI (right panel) of total Mo after administration of a single 60 mg ( $2 \times 30$ mg) dose of WTX101 uncoated capsules + PPI fasted to healthy | |
| | volunteers. | 15 |

# List of Abbreviations

| Term | Definition |
|---|---|
| λz | Elimination rate constant |
| AUC(0-t) | Area under the plasma concentration-time curve from 0 to the final time with a concentration $\geq$ LOQ. |
| AUC(inf) | Area under the plasma concentration-time curve to infinity |
| BMI | Body Mass Index |
| CL/F | Total clearance uncorrected for bioavailability (F) |
| cm | Centimeter |
| Cmax | Maximum plasma concentration |
| Cu | Copper |
| EC | Enteric coated |
| F | Bioavailability |
| h | hour |
| ICP-MS | Inductively coupled plasma mass spectrometry |
| kg | Kilogram |
| LOQ | Validated lower limit of the bioanalytical method(s) |
| m <sup>2</sup> | Meter Squares |
| mg | Milligram |
| mL | Milliliter |
| Mo | Molybdenum |
| MW | Molecular weight |
| ng | nanogram |
| PK | Pharmacokinetics |
| PPI | Proton Pump Inhibitor |
| QD | Once daily |
| r <sup>2</sup> | Coefficient of determination |
| t½ | Elimination half-life |
| Tlag | Absorption lag time |
| Tmax | Time of maximum plasma concentration |
| UC | Uncoated Capsule |
| Vz/F | Volume of distribution uncorrected for bioavailability (F) |

# 1.0 Synopsis of Pharmacokinetic Results

Protocol WTX101-102 was an open-label, 3-treatment, 3-period, 6-sequence, single-dose, randomized crossover study of the pharmacokinetics and comparative bioavailability of WTX101 after administration of an Enteric Coated (EC) Tablet versus dosing with the current uncoated capsule (UC) coadministered with a proton pump inhibitor (PPI; omeprazole) under fasting conditions and the effect of dosing an EC Tablet with and without food on the absorption of WTX101. Subjects received, according to a randomization schedule (Appendix I), 1 of the WTX101 treatments. Dosing occurred after an overnight fast (Treatments A and C) or 30 minutes after ingesting a high calorie / high fat meal (Treatment B) and there was a minimum 14-day washout between the dosing in successive periods.

Eighteen (18) subjects were enrolled into and completed the study. One (1) subject had a pre-dose plasma concentration after administration of the EC Tablet Fed that was  $\geq$  LOQ and  $\geq$  5% of the corresponding Cmax and was excluded from the descriptive statistics and statistical analyses for that treatment. The PK analysis population was therefore comprised of 18 subjects for the EC Tablet Fasted and the UC + PPI Fasted and 17 subjects for the EC Tablet Fed.

- Based on total Mo, administration of the EC Tablet Fasted results in comparable exposure to the UC + PPI Fasted in most subjects.
- Based on total Mo, administration of the EC Tablet Fed results in a 60% to 75% decrease in exposure compared to the EC Tablet Fasted in the majority of subjects.
- The mean  $t\frac{1}{2}$  for total Mo was essentially the same for all 3 treatments, with an overall mean of ~48 h or 2 days.
- There were no apparent relationships between CL/F and body size (weight, BMI), suggesting that a fixed dose, rather than a dose based on body size, i.e. mg/kg or mg/m², may be appropriate for WTX101.

- The lowest between-subject coefficients of variation (BSCV) for Cmax, AUC(0-t), and AUC(inf) were observed for the UC + PPI Fasted, with an ~2-fold increase when the EC Tablet was administered under fasted conditions and an ~4-fold increase, based on the AUCs, when the EC Tablet was administered under fed conditions.
- Administration of WTX101 either as the UC + PPI or the EC Tablet under fasted conditions should result in comparable plasma concentrations of total Mo in most subjects. However, administration of the EC Tablet under fed conditions results in a large decrease in exposure with increased between-subject variability.

#### 2.0 Introduction

WTX101 is an oral de-coppering agent. It is a bis-choline salt of tetrathiomolybdate, bis[(2-hydroxyethyl)trimethylammonium] tetrathiomolybdate. WTX101 is being developed by Wilson Therapeutics for the treatment of Wilson Disease (WD). WD is a rare autosomal-recessive disorder caused by mutations in the ATP7B gene, resulting in a disturbed copper (Cu) metabolism. In the affected patients, Cu accumulates in the liver and in other tissues including the central nervous system. Left untreated, morbidity is progressive and the condition is eventually fatal.

In previous studies, coadministration of proton pump inhibitors (PPI) has been shown to increase the bioavailability of tetrathiomolybdate and to reduce gastrointestinal side effects. An Enteric Coated (EC) tablet formulation would be expected to offer the same benefits of increased bioavailability and reduced gastrointestinal side effects while avoiding the need to coadminister a PPI.

This study was conducted as a crossover study, aimed at evaluating the absorption of WTX101 from the EC tablet under fed and fasted conditions and compared to the current uncoated capsule (UC) administered with a proton pump inhibitor (PPI; omeprazole) under fasting conditions.

#### 3.0 Objective

The primary objectives of the study were to evaluate:

- The effect of dosing with an EC tablet versus dosing with the current UC coadministered with a PPI under fasting conditions, on the absorption of WTX101.
- The effect of dosing an EC Tablet with and without food on the absorption of WTX101.
- The safety and tolerability of WTX101.

#### 4.0 Study Conduct

#### 4.1 Clinical

This study was conducted at Celerion, 621 Rose Street, Lincoln, NE 68502, under the direction of PPD

A copy of the protocol is included in the clinical summary that accompanies this report.

# 4.2 Bioanalytical

Plasma concentrations of total molybdenum (Mo) were measured using an Inductively coupled plasma mass spectrometry (ICP-MS) method by QPS Netherlands B.V., Petrus Campersingel 123, 9713 AG Groningen, The Netherlands. A detailed report of the bioanalytical methodology and results accompanies this report.

## 4.3 Pharmacokinetic and Statistical Analyses

The PK and statistical analyses were done by PPD Kramer Consulting LLC, 14313 Outpost Way, North Potomac, MD 20878, and are the subject of this report.

# 5.0 Overview of the Study Design

This was an open-label, 3-treatment, 3-period, 6-sequence, single-dose, randomized crossover study of the pharmacokinetics and comparative bioavailability of WTX101 after administration of an EC Tablet versus dosing with the current UC + PPI under fasting conditions and the effect of dosing an EC Tablet with and without food on the absorption of WTX101.

The treatments to be administered were as follows:

Treatment A: WTX101 EC Tablets, 60 mg (2 × 30 mg) at Hour 0 on Day 1 following an overnight fast.

Treatment B: WTX101 EC Tablets, 60 mg (2 × 30 mg) at Hour 0 on Day 1, 30 minutes after the start of a high-fat breakfast, preceded by an overnight fast.

Treatment C: WTX101 UC, 60 mg ( $2 \times 30$  mg), after an overnight fast, preceded by omeprazole 20 mg ( $1 \times 20$  mg delayed-release tablet) once-daily the mornings of Day -5 to Day -1.

Eighteen (18) healthy adult male and female volunteers were randomly assigned (Appendix I) to 1 of 6 treatment sequences, as shown in Table 1.

| | Treatment* | | |
|----------|------------|----------|----------|
| Sequence | Period 1 | Period 2 | Period 3 |
| 1 | A | В | C |
| 2 | В | C | A |
| 3 | С | A | В |
| 4 | В | A | C |
| 5 | A | C | В |
| 6 | C | D | ٨ |

Table 1: Treatment Sequences.

On Study Days 1, 15, and 29 (Periods 1, 2, and 3, respectively), blood samples for the determination of total Mo concentrations were collected before and at 1, 2, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, and 192 hours after dosing. Samples collected through 48 hours were on an inpatient basis and from 72 through 192 hours on an outpatient basis. There was a minimum 14-day washout between the dosing in each period.

#### 6.0 Pharmacokinetic and Statistical Methods

## 6.1 Pharmacokinetic Methods

All PK parameters were calculated using non-compartmental analysis. Only those plasma concentrations equal to or greater than the respective LOQ (total Mo –

<sup>\*</sup>A = WTX101 EC Tablets, 60 mg (2  $\times$  30 mg) fasted; B = WTX101 EC Tablets, 60 mg (2  $\times$  30 mg) fed; C = WTX101 UC 60 mg (2  $\times$  30 mg) + PPI fasted

0.1 ng/mL) were used in the analysis. Plasma concentrations < LOQ were taken as 0 for the calculation of the descriptive statistics for plasma concentrations at each sampling time. For the pharmacokinetic analysis, plasma concentrations < LOQ that occurred from pre-dose to the first concentration  $\geq$  LOQ were treated as 0 and those that occur thereafter were treated as missing. Actual sampling times were used for all pharmacokinetic analyses. Protocol times were used to calculate mean plasma concentrations for graphical displays.

The maximum plasma concentration (Cmax) and time to Cmax (Tmax) were taken directly from the data. If the plasma concentration at the 1<sup>st</sup> sample after drug administration — 1 h — was < LOQ, then the absorption lag time (Tlag) was taken as the 1<sup>st</sup> succeeding sampling time with a concentration  $\geq$  LOQ. The elimination rate constant,  $\lambda z$ , was calculated as the negative of the slope of the terminal log-linear segment of the plasma concentration-time curve. The slope was determined from a plot of the natural log of the terminal plasma concentrations against time; at least 3 terminal plasma concentration time points, beginning with the final concentration  $\geq$  LOQ, were selected for the determination of  $\lambda z$  and the regression will have a coefficient of determination (r<sup>2</sup>)  $\geq$  0.9000. The range of data used for each subject and treatment was determined by visual inspection of a semi-logarithmic plot of concentration vs. time. Elimination half-life (t½) was calculated according to the following equation.

$$t^{1/2} = \frac{0.693}{\lambda z}$$

Area under the curve from zero to the final sample with a concentration  $\geq$  LOQ [AUC(0-t)] was calculated using the linear trapezoidal method and extrapolated to infinity [AUC(inf)] using

$$AUC(\inf) = AUC(0-t) + \frac{C_{tf}}{\lambda z}$$

where  $C_{tf}$  is the final concentration  $\geq LOQ$ .

The clearance (CL/F) and volume of distribution (Vz/F) of Mo, uncorrected for bioavailability (F), were calculated according to

$$CL/F = \frac{Dose}{AUC(\inf)}$$
 and  $Vz/F = \frac{Dose}{AUC(\inf) \times \lambda z}$ ,

respectively, where Dose represents the dose of Mo. The molecular weights (MW) of WTX101 and Mo are 432.52 and 95.94, respectively, and thus 60 mg of WTX101 represents 13.3 mg of Mo.

All pharmacokinetic calculations were done and individual subject plasma concentration-time graphs were prepared using SAS<sup>®</sup> for Windows<sup>®</sup> Version 9.3. Graphs of mean plasma concentration vs. time and other in-text graphs were prepared using SigmaPlot for Windows Version 12.5.

## **6.2** Statistical Methods

Plasma concentrations, actual blood sampling times, and pharmacokinetic parameters are listed; concentrations and pharmacokinetic parameters are summarized using descriptive statistics.

All statistical analyses were done using SAS® for Windows® Version 9.3.

## 6.2.1 Primary Analysis

The PK parameters for total Mo — Cmax, AUC(0-t), and AUC(inf) — were compared between treatments using an Analysis of Variance (ANOVA) statistical model with sequence, treatment, and period as the fixed effects and subject within sequence as a random effect, using the natural logarithms of the data.

Confidence intervals (90%) were constructed for the least squares geometric mean ratios (GMR) — Treatment B (EC Tablet Fed)-to-Treatment A (EC Tablet Fasted) and Treatment A (EC tablet Fasted)-to-Treatment C (UC + PPI Fasted) — of all 3 parameters using the natural log-transformed data and the two one-sided t-tests procedure. The GMRs and associated 90% confidence limits (CI) were exponentiated back to the original scale.

## 6.2.2 Secondary Analysis

The within-subject coefficient of variation (WSCV) of Cmax, AUC(0-t), and AUC(inf) were estimated using

$$WSCV = 100\% \times \sqrt{e^{MSE} - 1}$$

where MSE is the mean squared error from the ANOVA.

## **6.2.3** Exploratory Analysis

Relationships between CL/F and body size — weight (kg) and BMI (kg/m² — were examined graphically for each treatment. If suggested by the graphs, regression models could be fit to the data.

#### 7.0 Results

The random code is shown in Appendix I and the individual subject body size — weight and body mass index (BMI) — are listed in Appendix II. The individual subject plasma total Mo concentrations, actual blood sampling times, and descriptive statistics for plasma concentrations are listed in Appendix III, Appendix IV, and Appendix V respectively. Individual subject PK parameters are listed in Appendix VI and the associated descriptive statistics for the PK parameters are in Appendix VII. The statistical analysis of the total Mo PK parameters is in Appendix VIII. Individual subject graphs of plasma total Mo concentration vs. time on linear axes can be found in Appendix IX and on semi-logarithmic axes in Appendix X. The latter contains line segments indicating the range of data used to estimate λz for those datasets for which it could be estimated.

## 7.1 Subjects with a Pre-Dose Concentration $\geq$ LOQ

Two (2) subjects had a plasma total Mo concentration prior to dosing in Period 2 that was ≥ LOQ (0.1 ng/mL) (Table 2). For Subject PPD the pre-dose concentration was 40.60% of the corresponding Cmax and the data for this treatment — EC Tablet Fed — for this subject was excluded from the descriptive statistics and statistical analyses. For Subject PPD the pre-dose concentration after administration of the UC + PPI Fasted was < 5% of

the corresponding Cmax (Table 2) and the data were therefore included in the descriptive statistics and the PK and statistical analyses.<sup>1</sup>

Table 2: Subjects with a pre-dose concentration  $\geq$  LOQ.

| Subject | Period | Treatment | C(0)<br>(ng/mL) | Cmax<br>(ng/mL) | Ratio*<br>(%) |
|---|---|---|---|---|---|
| PPD | 2 | EC Tablet Fed | 12.34 | 30.39 | 40.60 |
| | 2 | UC + PPI Fasted | 10.28 | 375.17 | 2.74 |

<sup>\*</sup>Ratios > 5% are shown in red.

Source: C(0) – Appendix III; Cmax – Appendix VI.

# 7.2 Pharmacokinetic Analysis Population

Eighteen (18) subjects were enrolled into and all completed the study. As discussed in Section 7.1, the data for Subject PPD for the EC Tablet Fed were excluded from the descriptive statistics and statistical analyses. The PK analysis population was therefore comprised of 18 subjects for the EC Tablet Fasted and the UC + PPI Fasted and 17 subjects for the EC Tablet Fed.

#### 7.3 Pharmacokinetics

#### **7.3.1** Results

The mean  $\pm$  standard error plasma concentrations of total Mo are shown in.

As shown in Figure 1, the mean ± standard error plasma concentrations of total Mo were slightly lower after administration of the EC Tablet Fasted compared to the UC + PPI Fasted. There was, however, variability among subjects with 3 of the 18 showing much lower concentrations for the EC Tablet, 5 showing the same pattern as the mean data, and 10 showing more comparable or superimposable concentrations for both treatments (Appendix IX).

Consistent with the mean plasma concentrations, the arithmetic (Table 3) and geometric (Table 4) mean values for Cmax, AUC(0-t), and AUC(inf) were lower for the EC Tablet Fasted than for the UC Capsule + PPI Fasted. The GMRs ranged from 75.81% to 87.16% with lower limits of the associated 90% CIs < 80.00% (Table 4), indicating a decrease in exposure *on the average*. The median Tmax was comparable for both

treatments, 4.54 h and 4.50 h, respectively, with comparable ranges (Table 3). Four (4) of the 18 subjects had an absorption lag time after administration of the EC Tablet fasted with a median (range) of 2.00 h (2.00 h to 3.00 h) (Table 3).

Administration of the EC Tablet with food resulted in a large decrease in the mean plasma total Mo concentrations (Figure 1). This was also observed in all but 2 of the 17 subjects evaluable for this treatment (Appendix IX). Cmax, AUC(0-t), and AUC(inf) were lower after administration of the EC Tablet with food (Table 3, Table 4) with GMRs ranging from 25.20% to 40.49%, indicating a substantial decrease in absorption. The median Tmax was comparable with and without food, 4.55 h and 4.54 h, respectively, with comparable ranges (Table 3). Compared to the EC Tablet Fasted, more subjects (6) had an absorption lag time an increase in the median (range) to 3.00 h (2.00 h to 5.00 h) (Table 3).

The mean  $t\frac{1}{2}$  was essentially the same for all 3 treatments (Table 3), with an overall mean of ~48 h or 2 days.

The relationships between Mo CL/F and body size, expressed as weight and BMI, are illustrated in Figure 2 (Treatment A — EC Tablet Fasted) and Figure 3 (Treatment C — UC + PPI Fasted). There are no apparent relationships between CL/F and either measure of body size. This suggests that a fixed dose, rather than a dose based on body size, i.e. mg/kg or mg/m², may be appropriate for WTX101.

The lowest between-subject coefficients of variation (BSCV) for Cmax, AUC(0-t), and AUC(inf) were observed for the UC capsule + PPI Fasted, with values ranging from 15.8% to 19.1% (Table 5). Administration of the EC Tablet Fasted resulted in higher BSCVs (26.1% to 35.2%; Table 5). The BSCVs were much higher, particularly for AUC(0-t) and AUC(inf) — 81.5% and 72.6%, respectively (Table 5) — when the EC Tablet was administered after the high calorie / high fat meal. Compared to the EC

\_

<sup>&</sup>lt;sup>1</sup> Due to the slight but apparent differences in bioavailability among the treatments, the relationships between CL/F and body size are shown separately for the 2 fasted treatments. As a consequence of the low bioavailability after administration of the EC Tablet Fed, it was excluded from this analysis.

Wilson Therapeutics USA, Inc. Study WTX101-102

Page 10 July 14, 2014

Tablet Fasted, the BSCVs for the AUCs were ~2.2-fold higher when the EC Tablet was administered under fed conditions.

Figure 1: Mean ± standard error plasma concentrations of total Mo after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC Tablets under fasted and fed conditions and UC + PPI under fasted conditions — linear axes (left panel) and semi-logarithmic (right panel).



Table 3: Summary of total Mo PK parameters after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC Tablets under fasted and fed conditions and UC + PPI under fasted conditions.

| | Treatment | | |
|---|---|---|---|
| Parameter* | EC Tablet Fasted | EC Tablet Fed | UC + PPI Fasted |
| Tlag (h) | 2.00 (4) | 3.00 (6) | — <del>†</del> |
| | [2.00 - 3.00] | [2.00 - 5.00] | |
| Cmax (ng/mL) | $376 \pm 98.0 (18)$ | $187 \pm 118 (17)$ | $442 \pm 69.6 (18)$ |
| Tmax (h) | 4.54 (18) | 4.55 (17) | 4.50 (18) |
| | [3.00 - 9.53] | [3.52 - 9.51] | [2.99 - 10.0] |
| $AUC(0-t) (h\times ng/mL)$ | $16,026 \pm 5,635 \ (18)$ | 5,740 ± 4,681 (17) | $19,809 \pm 3,509 (18)$ |
| $AUC(inf) (h \times ng/mL)$ | $17,258 \pm 5,955 (18)$ | $6,973 \pm 5,065 (15)$ | $21,047 \pm 4,022 \ (17)$ |
| $\lambda z (1/h)$ | $0.0140 \pm 0.0023$ (18) | $0.0258 \pm 0.0303$ (15) | $0.0145 \pm 0.0014$ (17) |
| t½ (h) | $51.0 \pm 8.87 (18)$ | $43.5 \pm 20.9 (15)$ | $48.2 \pm 4.86 (17)$ |
| CL/F (L/h) | $0.92 \pm 0.51 \ (18)$ | $6.34 \pm 11.9 (15)$ | $0.66 \pm 0.13$ (17) |
| Vz/F (L) | $66.6 \pm 34.0 (18)$ | $175 \pm 98.1 (15)$ | $45.2 \pm 8.31 (17)$ |

<sup>\*</sup>Arithmetic mean ± standard deviation (N) except for Tmax for which the median (N) [Range] is reported. Additional descriptive statistics can be found in Appendix VII.

Source: Appendix VII.

<sup>†</sup>Parameter could not be estimated for any subject for this treatment.

Table 4: Statistical analysis of total Mo PK parameters after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC Tablets under fasted and fed conditions and UC + PPI under fasted conditions.

| | Least Squares Geometric Means Geometric Mean Ratio (%)* | | | Within-Subject | |
|---|---|---|---|---|---|
| Parameter | Test | Reference | Estimate | 90% Confidence Inter | rval CV(%) |
| EC Tablet Fasted v | s. UC + PPI Fasted | | | | |
| Cmax | 360.88 | 436.61 | 82.65 | $63.91 \rightarrow 106$ | 5.90 47.98 |
| AUC(0-t) | 14,790.84 | 19,511.14 | 75.81 | 52.23 → 110 | 0.02 73.76 |
| AUC(inf) | 15,997.76 | 18,353.45 | 87.16 | 64.59 → 117 | 7.63 55.30 |
| EC Tablet Fed vs. l | <br>EC Tablet Fasted | | | | |
| Cmax | 146.11 | 360.88 | 40.49 | $31.12 \rightarrow 52$ | 2.68 47.98 |
| AUC(0-t) | 3,726.71 | 14,790.84 | 25.20 | $17.21 \rightarrow 36$ | 5.89 73.76 |
| AUC(inf) | 5,071.14 | 15,997.76 | 31.70 | $23.12 \rightarrow 43$ | 55.30 |

<sup>\*</sup>Based on analysis of natural log-transformed data.

Source: Appendix VIII.

Figure 2: Individual subject CL/F vs. body weight (left panel) and BMI (right panel) of total Mo after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC Tablets fasted to healthy volunteers.



Figure 3: Individual subject CL/F vs. body weight (left panel) and BMI (right panel) of total Mo after administration of a single 60 mg (2 × 30 mg) dose of WTX101 uncoated capsules + PPI fasted to healthy volunteers.



Table 5: Summary of between-subject coefficients of variation of total Mo Cmax, AUC(0-t), and AUC(inf) after administration of a single 60 mg (2 × 30 mg) dose of WTX101 EC Tablets under fasted and fed conditions and UC + PPI under fasted conditions.

| | Treatment | | |
|---|---|---|---|
| Parameter* | EC Tablet Fasted | EC Tablet Fed | UC + PPI Fasted |
| Cmax (ng/mL) | 26.1 | 39.9 | 15.8 |
| $AUC(0-t) (h \times ng/mL)$ | 35.2 | 81.5 | 17.7 |
| $AUC(inf) (h \times ng/mL)$ | 34.5 | 72.6 | 19.1 |

<sup>\*</sup>Between-subject coefficient of variation (%).

Source: Appendix VII.

## 7.3.2 Discussion

As illustrated in Figure 1, there was a slight decrease in the mean ± standard error plasma concentrations of total Mo after administration of the EC Tablet Fasted compared to the UC + PPI fasted. Similar trends were observed with respect to Cmax, AUC(0-t), and AUC(inf) (Table 3 and Table 4). Nevertheless, examination of the individual subject data (PK parameters — Appendix VI; graphs of plasma concentrations — Appendix IX) indicates that while a similar pattern was observed with some of the individual subjects, the majority had a total Mo concentration-time profile that was comparable for the EC Tablet and UC + PPI when both were administered under fasted conditions. However, administration of the EC Tablet fed resulted in a 60% to 75% decrease in absorption which was consistent among the majority of subjects (Appendix IX).

Administration of WTX101 as the EC Tablet increased the between-subject variability compared to the UC + PPI, ~2-fold when administered under fasted conditions and ~4-fold, based on the AUCs, when administered under fed conditions.

#### 8.0 Conclusions

- Based on total Mo, administration of the EC Tablet Fasted results in comparable exposure to the UC + PPI Fasted in most subjects.
- Based on total Mo, administration of the EC Tablet Fed results in a 60% to 75% decrease in exposure compared to the EC Tablet Fasted in the majority of subjects.
- The mean  $t\frac{1}{2}$  for total Mo was essentially the same for all 3 treatments, with an overall mean of ~48 h or 2 days.
- There were no apparent relationships between CL/F and body size (weight, BMI), suggesting that a fixed dose, rather than a dose based on body size, i.e. mg/kg or mg/m², may be appropriate for WTX101.
- The lowest between-subject coefficients of variation (BSCV) for Cmax, AUC(0-t), and AUC(inf) were observed for the UC + PPI Fasted, with an ~2-fold increase when

the EC Tablet was administered under fasted conditions and an ~4-fold increase, based on the AUCs, when the EC Tablet was administered under fed conditions.

 Administration of WTX101 either as the UC + PPI or the EC Tablet under fasted conditions should result in comparable plasma concentrations of total Mo in most subjects. However, administration of the EC Tablet under fed conditions results in a large decrease in exposure with increased between-subject variability.

## 9.0 References

Bioavailability and Bioequivalence Studies for Orally Administered Drug Products
 — General Considerations. U.S. Department of Health and Human Services, Food
 and Drug Administration, Center for Drug Evaluation and Research (CDER), March,
 2003.
Appendix I Random Code

| | | | — Treatment | |
|--------|------------|--------|-------------|--------|
| | | Period | Period | Period |
| Subjec | t Sequence | 1 | 2 | 3 |
| PPD | BCA | В | C | A |
| | BAC | В | A | C |
| | ABC | A | B | C |
| | CAB | C | A | В |
| | ACB | A | C | В |
| | CBA | C | В | A |
| | BCA | В | C | A |
| | ABC | A | В | С |
| | CBA | C | В | A |
| | CAB | C | A | В |
| | ACB | A | С | В |
| | BAC | В | A | С |
| | BAC | В | A | С |
| | CBA | С | В | A |
| | ABC | A | В | С |
| | BCA | В | С | A |
| | CAB | C | A | В |
| | ACB | A | С | В |

Treatment A - EC Tablet Fasted; Treatment B - EC Tablet Fed; Treatment C - Uncoated Capsule + PPI Fasted

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix II Subject Sex, Height, Weight, and BMI

| Subject | Sex | Height (cm)* | Weight<br>(kg)* | BMI<br>(kg/m²)§ |
|---------|-----|--------------|-----------------|-----------------|
| PPD | | 179 | 66.7 | 20.82 |
| | | 179 | 92.4 | 28.84 |
| | | 168 | 80.4 | 28.49 |
| | | 170 | 85.3 | 29.52 |
| | | 180 | 80.2 | 24.75 |
| | | 173 | 90.7 | 30.31 |
| | | 161 | 80.0 | 30.86 |
| | | 182 | 91.4 | 27.59 |
| | | 165 | 74.3 | 27.29 |
| | | 159 | 62.2 | 24.60 |
| | | 176 | 92.6 | 29.89 |
| | | 168 | 66.1 | 23.42 |
| | | 182 | 99.7 | 30.10 |
| | | 165 | 83.9 | 30.82 |
| | | 181 | 104.7 | 31.96 |
| | | 159 | 69.5 | 27.49 |
| | | 168 | 65.1 | 23.07 |
| | | 178 | 72.0 | 22.72 |

\*Screening values. \$Calculated from height and weight. Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix III Individual Subject Plasma Concentrations Treatment A - EC Tablet Fasted

| | | | | | | | s | cheduled | Time (h | .) ——— | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 0 | 1 | 2 | 3 | 3.5 | 4 | 4.5 | 5 | 6 | 7 | 7.5 | 8 | 8.5 | 9 |
| PPD | | | | | | | | | | | | | | | |
| | 3 | 0.00 | 98.18 | 125.71 | 138.32 | 134.78 | 134.68 | 147.29 | 144.71 | 127.97 | 115.04 | 116.83 | 112.36 | 117.64 | 105.05 |
| | 2 | 0.00 | 131.56 | 181.29 | 254.30 | 259.03 | 265.79 | 259.69 | 236.91 | 232.83 | 236.22 | 249.49 | 258.13 | 269.11 | 261.36 |
| | 1 | 0.00 | 103.85 | 123.14 | 201.11 | 228.55 | 235.67 | 278.51 | 254.12 | 233.12 | 222.06 | 218.52 | 208.76 | 211.79 | 210.42 |
| | 2 | 0.00 | 216.94 | 291.58 | 441.89 | 426.36 | 384.91 | 386.73 | 359.17 | 343.18 | 348.62 | 329.94 | 328.22 | 314.16 | 314.27 |
| | 1 | 0.00 | 0.00 | 0.00 | 137.20 | 178.68 | 193.81 | 264.12 | 256.91 | 361.37 | 391.14 | 397.87 | 390.01 | 349.42 | 366.02 |
| | 3 | 0.00 | 51.16 | 230.61 | 322.23 | 381.35 | 396.83 | 450.27 | 407.18 | 395.63 | 430.82 | 417.64 | 441.73 | 420.96 | 416.72 |
| | 3 | 0.00 | 34.22 | 218.85 | 366.40 | 401.36 | 399.91 | 445.21 | 434.97 | 459.26 | 466.89 | 471.67 | 460.54 | 443.90 | 406.51 |
| | 1 | 0.00 | 103.97 | 215.77 | 372.46 | 411.20 | 361.31 | 393.54 | 339.88 | 335.44 | 342.55 | 335.99 | 340.47 | 338.79 | 350.50 |
| | 3 | 0.00 | 0.00 | 176.32 | 250.96 | 285.75 | 323.16 | 378.18 | 421.52 | 450.94 | 422.34 | 419.15 | 410.65 | 384.26 | 396.16 |
| | 2 | 0.00 | 126.94 | 224.27 | 325.68 | 389.12 | 407.87 | 424.72 | 377.99 | 345.06 | 340.38 | 350.33 | 350.58 | 347.63 | 346.22 |
| | 1 | 0.00 | 85.14 | 207.71 | 291.54 | 329.85 | 325.93 | 362.73 | 359.79 | 333.19 | 350.12 | 342.13 | 345.30 | 346.02 | 363.13 |
| | 2 | 0.00 | 47.05 | 284.76 | 348.80 | 429.67 | 445.57 | 445.60 | 392.73 | 363.19 | 352.16 | 346.38 | 364.62 | 361.13 | 345.61 |
| | 2 | 0.00 | 131.22 | 232.84 | 309.63 | 288.91 | 283.82 | 337.12 | 313.26 | 295.05 | 268.31 | 272.14 | 301.30 | 293.73 | 328.17 |
| | 3 | 0.00 | 164.45 | 281.99 | 344.07 | 366.83 | 392.60 | 349.50 | 317.17 | 313.08 | 295.65 | 312.10 | 314.15 | 288.54 | 308.53 |
| | 1 | 0.00 | 41.02 | 58.40 | 56.51 | 62.06 | 121.48 | 185.29 | 226.50 | 355.54 | 296.63 | 297.73 | 296.64 | 277.83 | 292.64 |
| | 3 | 0.00 | 0.00 | 51.89 | 143.01 | 145.26 | 166.39 | 213.74 | 212.31 | 218.93 | 217.18 | 219.93 | 198.39 | 207.42 | 205.77 |
| | 2 | 0.00 | 137.79 | 182.76 | 224.62 | 252.50 | 271.86 | 312.57 | 298.54 | 298.64 | 289.98 | 286.18 | 279.42 | 273.04 | 268.70 |
| | 1 | 0.00 | 0.00 | 195.53 | 337.83 | 413.32 | 478.14 | 533.87 | 483.43 | 483.92 | 461.07 | 460.39 | 464.76 | 484.69 | 467.48 |

 $\label{eq:assaylog} Assay \ \mbox{LOQ} = 10 \ \mbox{ng/mL} \\ \mbox{(. = no sample analyzed and/or reported)}$ 

Wilson Therapeutics USA, Inc.
Study WTX101-102
July 14, 2014

Appendix III Individual Subject Plasma Concentrations Treatment A - EC Tablet Fasted

| | | | | | | | S | cheduled | Time (h | 1) ——— | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 9.5 | 10 | 12 | 14 | 16 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | 192 |
| PPD | | | | | | | | | | | | | | | |
| PPD | 3 | 112.76 | 99.92 | 95.51 | 88.90 | 79.60 | 60.92 | 47.59 | 35.30 | 21.94 | 14.71 | 10.78 | 0.00 | 0.00 | 0.00 |
| | 2 | 260.79 | 236.14 | 227.19 | 204.69 | 185.09 | 147.11 | 107.47 | 82.48 | 50.55 | 33.55 | 22.31 | 16.23 | 12.86 | 0.00 |
| | 1 | 225.06 | 205.92 | 176.43 | 157.93 | 152.88 | 97.47 | 69.32 | 51.19 | 30.31 | 17.98 | 12.76 | 0.00 | 0.00 | 0.00 |
| | 2 | 304.71 | 319.67 | 285.85 | 255.60 | 259.52 | 192.44 | 142.28 | 110.57 | 67.51 | 44.77 | 32.70 | 23.54 | 16.08 | 14.88 |
| | 1 | 352.32 | 348.76 | 335.61 | 316.58 | 294.79 | 225.15 | 173.69 | 129.75 | 93.38 | 63.95 | 47.64 | 32.45 | 22.88 | 17.83 |
| | 3 | 430.28 | 386.82 | 365.13 | 309.13 | 300.81 | 241.06 | 184.14 | 153.41 | 115.16 | 82.92 | 65.42 | 48.90 | 36.43 | 29.78 |
| | 3 | 483.93 | 439.16 | 412.80 | 380.54 | 356.82 | 278.09 | 197.75 | 165.38 | 109.70 | 71.94 | 48.97 | 35.21 | 26.33 | 21.32 |
| | 1 | 355.05 | 318.66 | 307.43 | 284.51 | 268.49 | 217.31 | 179.06 | 143.01 | 103.58 | 64.34 | 43.22 | 32.54 | 21.89 | 15.20 |
| | 3 | 402.79 | 381.36 | 343.25 | 336.71 | 312.59 | 229.49 | 170.57 | 139.00 | 83.68 | 56.87 | 38.65 | 25.64 | 19.56 | 14.94 |
| | 2 | 336.90 | 322.15 | 306.96 | 257.42 | 249.45 | 195.73 | 142.86 | 104.51 | 66.33 | 49.72 | 37.37 | 30.10 | 23.43 | 19.41 |
| | 1 | 382.79 | 339.11 | 336.56 | 305.76 | 284.98 | 218.45 | 176.12 | 142.62 | 94.04 | 69.13 | 48.73 | 36.28 | 27.56 | 23.57 |
| | 2 | 359.32 | 337.47 | 337.98 | 301.69 | 289.11 | 214.49 | 175.84 | 142.55 | 85.27 | 59.90 | 37.70 | 28.21 | 20.62 | 15.45 |
| | 2 | 370.37 | 353.17 | 322.89 | 323.13 | 300.35 | 232.70 | 184.84 | 148.69 | 95.31 | 63.80 | 47.80 | 32.00 | 26.70 | 19.35 |
| | 3 | 293.83 | 282.71 | 253.88 | 236.86 | 215.28 | 171.24 | 128.20 | 93.85 | 54.15 | 38.16 | 27.71 | 18.25 | 16.10 | 13.73 |
| | 1 | 283.95 | 262.86 | 235.97 | 217.67 | 179.96 | 139.98 | 108.75 | 80.09 | 49.45 | 31.58 | 24.04 | 17.77 | 14.03 | 10.97 |
| | 3 | 210.84 | 187.51 | 161.23 | 143.24 | 127.83 | 88.49 | 59.00 | 40.87 | 24.61 | 16.68 | 13.42 | 10.12 | 0.00 | 0.00 |
| | 2 | 288.20 | 266.03 | 263.01 | 249.57 | 231.03 | 170.63 | 135.96 | 115.92 | 72.60 | 47.06 | 37.47 | 27.27 | 21.64 | 15.26 |
| | 1 | 471.19 | 445.84 | 441.49 | 397.88 | 371.79 | 294.46 | 217.24 | 177.90 | 115.12 | 78.30 | 52.94 | 37.19 | 27.53 | 21.02 |

Assay LOQ = 10 ng/mL (. = no sample analyzed and/or reported)

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix III
Individual Subject Plasma Concentrations
Treatment B - EC Tablet Fed

| | | | | | | | S | cheduled | Time (h | .) ——— | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 0 | 1 | 2 | 3 | 3.5 | 4 | 4.5 | 5 | 6 | 7 | 7.5 | 8 | 8.5 | 9 |
| PPD | | | | | | | | | | | | | | | |
| FFD | 1 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 12.85 | 21.31 | 26.61 | 27.15 | 26.70 | 24.40 | 23.84 |
| | 1 | 0.00 | 0.00 | 19.53 | 73.01 | 103.86 | 122.75 | 144.33 | 144.19 | 136.16 | 125.60 | 124.38 | 118.22 | 112.11 | 109.29 |
| | 2 | 0.00 | 0.00 | 0.00 | 55.41 | 64.64 | 62.62 | 71.48 | 63.85 | 63.03 | 63.23 | 64.01 | 60.00 | 63.17 | 59.68 |
| | 3 | 0.00 | 17.63 | 163.84 | 295.07 | 338.70 | 365.88 | 386.35 | 369.95 | 362.28 | 355.71 | 357.16 | 362.04 | 351.14 | 361.03 |
| | 3 | 0.00 | 18.50 | 31.04 | 40.99 | 50.52 | 55.02 | 64.10 | 64.88 | 69.05 | 75.27 | 73.47 | 69.96 | 67.68 | 64.73 |
| | 2 | 12.34 | 11.91 | 11.82 | 16.32 | 18.79 | 20.68 | 24.66 | 26.31 | 27.81 | 29.98 | 30.06 | 30.39 | 29.06 | 29.90 |
| | 1 | 0.00 | 10.56 | 10.90 | 14.69 | 17.40 | 21.24 | 29.16 | 33.80 | 41.03 | 45.72 | 45.31 | 44.84 | 44.00 | 42.00 |
| | 2 | 0.00 | 100.70 | 223.00 | 270.10 | 278.69 | 250.68 | 246.98 | 224.48 | 203.37 | 186.22 | 177.73 | 170.61 | 172.76 | 163.03 |
| | 2 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 41.25 | 152.93 | 264.01 | 313.69 | 315.30 | 303.47 | 293.78 |
| | 3 | 0.00 | 0.00 | 69.44 | 155.16 | 180.68 | 214.36 | 231.05 | 226.73 | 247.67 | 250.60 | 228.21 | 235.55 | 231.30 | 213.13 |
| | 3 | 0.00 | 12.76 | 60.13 | 65.00 | 68.49 | 68.42 | 72.27 | 69.50 | 73.25 | 67.49 | 68.82 | 65.18 | 61.54 | 61.15 |
| | 1 | 0.00 | 0.00 | 0.00 | 95.61 | 269.48 | 294.17 | 314.87 | 298.13 | 290.46 | 298.33 | 265.11 | 265.05 | 236.01 | 264.11 |
| | 1 | 0.00 | 93.68 | 185.96 | 206.87 | 224.37 | 240.28 | 256.51 | 249.79 | 234.39 | 215.20 | 196.05 | 200.88 | 183.31 | 187.43 |
| | 2 | 0.00 | 122.88 | 116.09 | 123.52 | 127.48 | 125.11 | 137.05 | 130.62 | 120.55 | 120.76 | 114.42 | 121.14 | 112.86 | 118.34 |
| | 2 | 0.00 | 43.93 | 71.15 | 74.60 | 81.63 | 79.24 | 87.43 | 81.91 | 75.72 | 72.43 | 69.18 | 65.51 | 66.65 | 64.04 |
| | 1 | 0.00 | 63.64 | 174.22 | 232.66 | 264.35 | 262.92 | 272.07 | 264.48 | 257.48 | 228.43 | 234.69 | 218.01 | 208.02 | 202.39 |
| | 3 | 0.00 | 34.52 | 62.27 | 81.62 | 84.74 | 93.57 | 99.11 | 101.54 | 100.88 | 108.85 | 106.91 | 102.02 | 95.32 | 96.57 |
| | 3 | 0.00 | 48.89 | 176.75 | 273.72 | 293.40 | 309.80 | 325.45 | 298.39 | 290.22 | 270.46 | 254.53 | 258.93 | 244.79 | 238.98 |

 $\label{eq:assaylog} Assay \ \mbox{LOQ} = 10 \ \mbox{ng/mL} \\ \mbox{(. = no sample analyzed and/or reported)}$ 

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix III
Individual Subject Plasma Concentrations
Treatment B - EC Tablet Fed

| | | | | | | | S | Scheduled | l Time (h | ) ——— | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 9.5 | 10 | 12 | 14 | 16 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | 192 |
| PPD | | | | | | | | | | | | | | | |
| 110 | 1 | 22.74 | 20.35 | 15.83 | 12.49 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |
| | 1 | 102.40 | 93.88 | 83.54 | 70.40 | 58.36 | 41.73 | 28.68 | 20.40 | 12.26 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |
| | 2 | 61.95 | 54.64 | 44.48 | 40.03 | 36.43 | 27.97 | 14.59 | 11.88 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |
| | 3 | 387.75 | 361.80 | 336.48 | 287.92 | 271.27 | 205.55 | 164.40 | 123.25 | 81.51 | 46.99 | 31.11 | 22.42 | 16.87 | 14.10 |
| | 3 | 62.74 | 58.63 | 44.76 | 36.19 | 31.43 | 19.73 | 13.19 | 12.01 | 11.41 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |
| | 2 | 29.11 | 29.40 | 27.63 | 25.66 | 23.05 | 20.66 | 17.83 | 16.93 | 14.94 | 13.13 | 12.08 | 10.85 | 10.26 | 0.00 |
| | 1 | 40.88 | 38.50 | 31.95 | 25.93 | 22.45 | 15.08 | 10.09 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |
| | 2 | 144.14 | 150.50 | 129.38 | 116.44 | 104.83 | 77.62 | 56.59 | 44.71 | 33.05 | 20.90 | 16.58 | 12.05 | 11.52 | 0.00 |
| | 2 | 282.58 | 266.41 | 253.46 | 220.59 | 198.89 | 148.90 | 111.04 | 87.57 | 53.12 | 32.67 | 27.06 | 20.49 | 14.68 | 14.61 |
| | 3 | 209.67 | 197.77 | 166.45 | 161.87 | 135.22 | 99.25 | 73.16 | 49.52 | 34.18 | 27.16 | 20.07 | 14.23 | 12.49 | 11.45 |
| | 3 | 59.32 | 54.39 | 51.61 | 47.20 | 40.48 | 33.12 | 22.31 | 19.44 | 14.26 | 11.45 | 11.03 | 0.00 | 0.00 | 0.00 |
| | 1 | 243.44 | 217.27 | 206.65 | 202.29 | 168.90 | 124.03 | 88.83 | 70.95 | 40.85 | 26.10 | 19.04 | 12.84 | 10.08 | 0.00 |
| | 1 | 184.59 | 164.35 | 151.38 | 133.58 | 114.28 | 81.36 | 60.24 | 45.75 | 27.43 | 20.26 | 14.02 | 10.87 | 0.00 | 0.00 |
| | 2 | 119.70 | 112.78 | 104.55 | 95.49 | 83.22 | 59.42 | 36.81 | 28.19 | 17.43 | 12.95 | 0.00 | 0.00 | 0.00 | 0.00 |
| | 2 | 63.03 | 53.90 | 47.35 | 42.35 | 38.05 | 24.95 | 15.97 | 13.13 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 | 0.00 |
| | 1 | 214.18 | 193.12 | 165.25 | 148.12 | 122.52 | 86.84 | 53.00 | 39.10 | 22.72 | 16.69 | 12.37 | 0.00 | 0.00 | 0.00 |
| | 3 | 95.97 | 87.71 | 70.99 | 58.05 | 48.75 | 33.42 | 22.46 | 20.53 | 15.56 | 11.45 | 10.51 | 0.00 | 0.00 | 0.00 |
| | 3 | 241.80 | 217.08 | 199.77 | 170.73 | 155.83 | 118.87 | 82.46 | 60.69 | 42.21 | 29.73 | 22.87 | 17.90 | 15.04 | 12.28 |

Assay LOQ = 10 ng/mL (. = no sample analyzed and/or reported)

Appendix III
Individual Subject Plasma Concentrations
Treatment C - Uncoated Capsule + PPI Fasted

| | | | | | | | S | cheduled | l Time (h | .) ——— | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 0 | 1 | 2 | 3 | 3.5 | 4 | 4.5 | 5 | 6 | 7 | 7.5 | 8 | 8.5 | 9 |
| PPD | | | | | | | | | | | | | | | |
| PPD | 2 | 0.00 | 224.42 | 321.57 | 445.77 | 415.87 | 396.83 | 438.76 | 395.75 | 384.80 | 374.79 | 372.45 | 347.23 | 374.22 | 356.89 |
| | 3 | 0.00 | 192.87 | 226.09 | 306.50 | 353.87 | 320.33 | 313.55 | 293.74 | 303.75 | 302.48 | 291.78 | 296.67 | 303.73 | 303.22 |
| | 3 | 0.00 | 191.87 | 283.68 | 347.63 | 351.11 | 377.14 | 447.08 | 416.43 | 397.65 | 383.91 | 363.62 | 352.14 | 366.16 | 347.99 |
| | 1 | 0.00 | 177.57 | 327.32 | 409.25 | 399.03 | 418.87 | 460.34 | 386.95 | 375.68 | 381.60 | 356.53 | 374.77 | 378.81 | 367.19 |
| | 2 | 0.00 | 292.36 | 344.86 | 361.71 | 347.34 | 349.25 | 366.44 | 390.67 | 392.11 | 375.63 | 393.39 | 403.71 | 398.74 | 402.12 |
| | 1 | 0.00 | 146.44 | 297.86 | 371.24 | 367.63 | 392.13 | 402.97 | 375.76 | 394.88 | 376.46 | 383.51 | 388.41 | 393.68 | 381.60 |
| | 2 | 0.00 | 187.04 | 278.25 | 391.55 | 411.06 | 417.43 | 459.34 | 433.49 | 416.44 | 417.04 | 410.70 | 400.32 | 402.69 | 403.65 |
| | 3 | 0.00 | 172.51 | 302.15 | 346.64 | 366.56 | 359.30 | 367.72 | 327.67 | 327.51 | 320.73 | 303.08 | 300.30 | 304.80 | 299.41 |
| | 1 | 0.00 | 284.76 | 414.18 | 444.73 | 477.57 | 439.41 | 445.33 | 408.90 | 406.91 | 398.53 | 388.18 | 385.06 | 381.33 | 386.98 |
| | 1 | 0.00 | 217.16 | 347.86 | 421.06 | 422.30 | 504.29 | 566.16 | 508.98 | 494.04 | 484.56 | 453.48 | 454.36 | 462.01 | 460.35 |
| | 2 | 10.28 | 127.23 | 233.36 | 300.54 | 317.84 | 318.92 | 353.98 | 375.17 | 343.82 | 347.99 | 330.78 | 337.38 | 332.99 | 314.67 |
| | 3 | 0.00 | 238.80 | 391.08 | 496.93 | 456.00 | 405.66 | 403.10 | 354.45 | 341.59 | 332.72 | 335.86 | 356.96 | 386.74 | 369.44 |
| | 3 | 0.00 | 178.85 | 238.61 | 261.60 | 313.19 | 405.34 | 378.42 | 354.16 | 335.74 | 343.32 | 331.76 | 360.85 | 338.15 | 341.49 |
| | 1 | 0.00 | 229.28 | 307.83 | 378.54 | 423.01 | 514.24 | 567.10 | 511.19 | 455.47 | 445.27 | 460.56 | 434.12 | 452.59 | 433.62 |
| | 3 | 0.00 | 243.79 | 263.93 | 343.30 | 356.25 | 351.84 | 396.79 | 395.00 | 383.28 | 379.15 | 406.78 | 368.15 | 386.99 | 406.89 |
| | 2 | 0.00 | 244.56 | 331.66 | 430.38 | 525.94 | 487.14 | 506.36 | 522.42 | 500.18 | 466.81 | 490.01 | 457.84 | 466.42 | 469.08 |
| | 1 | 0.00 | 177.70 | 226.93 | 274.26 | 281.36 | 286.07 | 313.14 | 285.64 | 278.19 | 281.49 | 303.36 | 296.99 | 288.49 | 283.64 |
| | 2 | 0.00 | 214.52 | 303.38 | 375.11 | 434.78 | 460.50 | 460.65 | 389.43 | 389.19 | 384.06 | 384.60 | 392.86 | 392.85 | 387.66 |

 $\label{eq:assaylog} Assay \ \mbox{LOQ} = 10 \ \mbox{ng/mL} \\ \mbox{(. = no sample analyzed and/or reported)}$ 

Wilson Therapeutics USA, Inc.
Study WTX101-102
July 14, 2014

Appendix III
Individual Subject Plasma Concentrations
Treatment C - Uncoated Capsule + PPI Fasted

| | | | | | | | S | cheduled | Time (h | .) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 9.5 | 10 | 12 | 14 | 16 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | 192 |
| PPD | | | | | | | | | | | | | | | |
| PPD | 2 | 378.12 | 340.38 | 329.38 | 307.77 | 300.02 | 227.34 | 182.73 | 136.12 | 96.11 | 59.37 | 39.66 | 84.79 | 21.57 | 13.58 |
| | 3 | 304.27 | 276.50 | 273.22 | 237.39 | 221.39 | 168.44 | 134.43 | 95.76 | 56.85 | 35.40 | 24.03 | 16.75 | 12.92 | 10.21 |
| | 3 | 375.62 | 333.90 | 311.55 | 266.46 | 254.40 | 191.91 | 139.42 | 113.03 | 70.17 | 42.16 | 30.55 | 18.82 | 15.27 | 11.38 |
| | 1 | 380.14 | 360.12 | 352.32 | 319.54 | 283.43 | 216.70 | 160.60 | 123.93 | 77.34 | 49.76 | 33.11 | 21.40 | 15.51 | 12.34 |
| | 2 | 387.36 | 420.63 | 400.83 | 371.53 | 354.52 | 282.20 | 210.81 | 177.45 | 125.29 | 86.81 | 66.86 | 49.56 | 36.86 | 28.30 |
| | 1 | 377.46 | 368.36 | 346.78 | 314.09 | 296.17 | 244.65 | 184.02 | 156.60 | 116.31 | 82.97 | 55.69 | 45.11 | 36.09 | 27.35 |
| | 2 | 424.07 | 374.84 | 345.94 | 312.07 | 295.06 | 243.41 | 180.78 | 140.31 | 88.17 | 59.81 | 42.41 | 29.24 | 23.50 | 17.56 |
| | 3 | 312.16 | 276.55 | 257.41 | 245.59 | 227.29 | 178.21 | 146.10 | 112.61 | 73.32 | 47.69 | 36.56 | 25.66 | 18.57 | 14.14 |
| | 1 | 397.37 | 381.58 | 356.53 | 325.10 | 310.16 | 242.30 | 195.76 | 155.76 | 100.31 | 66.04 | 45.65 | 34.75 | 27.27 | 18.52 |
| | 1 | 476.75 | 475.05 | 483.18 | 444.36 | 411.71 | 331.55 | 248.04 | 191.50 | 123.79 | 86.90 | 60.70 | 45.69 | 35.64 | 27.27 |
| | 2 | 341.95 | 331.05 | 310.17 | 306.04 | 280.37 | 222.50 | 169.94 | 137.93 | 89.31 | 65.79 | 43.28 | 36.66 | 29.13 | 20.96 |
| | 3 | 371.57 | 362.27 | 326.69 | 303.20 | 273.45 | 217.46 | 179.13 | 132.44 | 87.33 | 51.20 | 36.17 | 26.28 | 19.93 | 13.58 |
| | 3 | 342.72 | 331.49 | 323.28 | 292.50 | 285.39 | 226.62 | 189.29 | 150.77 | 106.33 | 73.72 | 51.86 | 37.92 | 30.21 | 22.81 |
| | 1 | 425.94 | 411.98 | 383.88 | 339.51 | 300.50 | 227.74 | 171.68 | 125.20 | 82.82 | 54.73 | 36.22 | 26.31 | 21.26 | 17.41 |
| | 3 | 371.30 | 362.04 | 349.01 | 289.32 | 269.58 | 212.02 | 166.18 | 127.70 | 85.14 | 59.30 | 41.62 | 30.95 | 22.13 | 16.00 |
| | 2 | 479.68 | 447.22 | 399.67 | 423.13 | 370.26 | 278.32 | 208.34 | 156.94 | 102.21 | 67.16 | 45.48 | 32.12 | 25.40 | 21.03 |
| | 1 | 289.70 | 273.28 | 251.68 | 227.71 | 210.72 | 158.07 | 128.40 | 107.16 | 69.18 | 42.79 | 31.00 | 22.05 | 15.82 | 13.40 |
| | 2 | 427.60 | 411.21 | 373.99 | 342.50 | 315.24 | 262.80 | 197.64 | 160.18 | 108.44 | 76.12 | 51.59 | 38.53 | 28.04 | 20.71 |

 $\label{eq:assaylog} Assay \ \mbox{LOQ} = 10 \ \mbox{ng/mL} \\ \mbox{(. = no sample analyzed and/or reported)}$ 

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix IV
Individual Subject Blood Sampling Times
Treatment A - EC Tablet Fasted

| | | | | | | | S | cheduled | Time (h) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 0 | 1 | 2 | 3 | 3.5 | 4 | 4.5 | 5 | 6 | 7 | 7.5 | 8 | 8.5 | 9 |
| PPD | | | | | | | | | | | | | | | |
| | 3 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 2 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 1 | -0.66 | 1.00 | 2.00 | 3.00 | 3.51 | 4.01 | 4.50 | 5.00 | 6.01 | 7.00 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 2 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.02 | 7.50 | 8.00 | 8.50 | 9.01 |
| | 1 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.52 | 9.00 |
| | 3 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.03 | 8.51 | 9.00 |
| | 3 | -0.74 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 1 | -0.75 | 1.00 | 2.00 | 3.00 | 3.52 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.01 | 8.50 | 9.00 |
| | 3 | -0.75 | 1.00 | 2.00 | 3.01 | 3.50 | 4.00 | 4.52 | 5.00 | 6.00 | 7.02 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 2 | -0.53 | 1.01 | 2.12 | 3.01 | 3.52 | 4.00 | 4.55 | 5.01 | 6.00 | 7.01 | 7.51 | 8.11 | 8.55 | 9.01 |
| | 1 | -0.74 | 1.00 | 2.00 | 3.04 | 3.52 | 4.04 | 4.52 | 5.00 | 6.00 | 7.00 | 7.50 | 8.02 | 8.56 | 9.01 |
| | 2 | -0.73 | 1.01 | 2.01 | 3.01 | 3.53 | 4.00 | 4.53 | 5.00 | 6.00 | 7.01 | 7.51 | 8.01 | 8.51 | 9.00 |
| | 2 | -0.73 | 1.01 | 2.01 | 3.01 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.01 | 7.52 | 8.01 | 8.51 | 9.03 |
| | 3 | -0.75 | 1.09 | 2.01 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.52 | 8.01 | 8.51 | 9.01 |
| | 1 | -0.75 | 1.00 | 2.00 | 3.00 | 3.52 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.03 | 8.51 | 9.01 |
| | 3 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.52 | 8.01 | 8.52 | 9.02 |
| | 2 | -0.72 | 1.03 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.03 | 8.50 | 9.01 |
| | 1 | -0.75 | 1.00 | 2.00 | 3.00 | 3.51 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.01 | 8.51 | 9.00 |
| | _ | 0.75 | ± .00 | 2.00 | 5.00 | J.JI | 1.00 | 1.50 | 5.00 | 0.00 | , . 00 | , . 50 | 0.01 | 0.51 | 5.00 |

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix IV
Individual Subject Blood Sampling Times
Treatment A - EC Tablet Fasted

| | | | | | | | S | cheduled | Time (h) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 9.5 | 10 | 12 | 14 | 16 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | 192 |
| PPD | | | | | | | | | | | | | | | |
| ווט | 3 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.00 | 12.14 | 14.00 | 16.00 | 24.01 | 36.00 | 48.06 | 72.00 | 96.00 | 120.09 | 144.00 | 168.00 | 192.00 |
| | 1 | 9.52 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.01 | 48.00 | 72.01 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.01 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.01 | 72.00 | 96.01 | 120.09 | 144.01 | 168.01 | 192.01 |
| | 1 | 9.52 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.02 | 48.07 | 72.00 | 96.00 | 120.00 | 144.00 | 168.01 | 192.00 |
| | 3 | 9.50 | 10.00 | 12.00 | 14.05 | 16.00 | 24.00 | 36.05 | 48.00 | 72.00 | 96.00 | 120.01 | 144.00 | 168.00 | 192.00 |
| | 3 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 1 | 9.52 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.03 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 3 | 9.50 | 10.00 | 12.01 | 14.00 | 16.00 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.01 | 12.01 | 14.01 | 16.01 | 24.05 | 36.07 | 48.11 | 72.03 | 96.07 | 120.09 | 144.00 | 168.08 | 192.51 |
| | 1 | 9.53 | 10.01 | 12.00 | 14.02 | 16.03 | 24.01 | 36.06 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.01 | 192.00 |
| | 2 | 9.50 | 10.00 | 12.02 | 14.01 | 16.00 | 24.01 | 36.02 | 48.01 | 72.01 | 96.02 | 120.09 | 144.00 | 168.01 | 192.03 |
| | 2 | 9.51 | 10.03 | 12.03 | 14.01 | 16.00 | 24.01 | 36.01 | 48.01 | 72.01 | 96.02 | 120.09 | 144.00 | 168.01 | 192.03 |
| | 3 | 9.50 | 10.01 | 12.00 | 14.00 | 16.01 | 24.02 | 36.08 | 48.00 | 72.01 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 1 | 9.53 | 10.01 | 12.00 | 14.02 | 16.02 | 24.00 | 36.00 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.01 | 192.01 |
| | 3 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.01 | 36.10 | 48.00 | 72.01 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.51 | 10.01 | 12.15 | 14.01 | 16.00 | 24.04 | 36.02 | 48.03 | 72.01 | 96.02 | 120.10 | 144.00 | 168.01 | 192.03 |
| | 1 | 9.53 | 10.00 | 12.00 | 14.02 | 16.01 | 24.00 | 36.10 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.03 | 192.00 |

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix IV
Individual Subject Blood Sampling Times
Treatment B - EC Tablet Fed

| PPD 1 -0.75 1.00 2.00 3.00 3.50 4.00 4.50 5.00 6.00 7.00 7.50 1 -0.75 1.00 2.00 3.00 3.51 4.00 4.50 5.00 6.01 7.00 7.50 2 -0.71 1.00 2.01 3.00 3.50 4.00 4.50 5.00 6.00 7.02 7.50 3 -0.75 1.01 2.01 3.01 3.50 4.01 4.51 5.00 6.00 7.02 7.50 | | | |
|---|---|---|---|
| 1 -0.75 1.00 2.00 3.00 3.50 4.00 4.50 5.00 6.00 7.00 7.50<br>1 -0.75 1.00 2.00 3.00 3.51 4.00 4.50 5.00 6.01 7.00 7.50<br>2 -0.71 1.00 2.01 3.00 3.50 4.00 4.50 5.00 6.00 7.02 7.50 | 8 | 8.5 | 9 |
| 1 -0.75 1.00 2.00 3.00 3.50 4.00 4.50 5.00 6.00 7.00 7.50<br>1 -0.75 1.00 2.00 3.00 3.51 4.00 4.50 5.00 6.01 7.00 7.50<br>2 -0.71 1.00 2.01 3.00 3.50 4.00 4.50 5.00 6.00 7.02 7.50 | | | |
| 2 -0.71 1.00 2.01 3.00 3.50 4.00 4.50 5.00 6.00 7.02 7.50 | 8.00 | 8.50 | 9.00 |
| | 8.00 | 8.50 | 9.00 |
| 3 -0.75 1.01 2.01 3.01 3.50 4.01 4.51 5.00 6.00 7.00 7.50 | 8.01 | 8.50 | 9.01 |
| 0 01/0 21/02 01/02 01/02 11/02 01/00 01/00 71/00 | 8.01 | 8.50 | 9.00 |
| 3 -0.75 1.01 2.01 3.01 3.50 4.00 4.50 5.00 6.00 7.00 7.50 | 8.01 | 8.50 | 9.00 |
| 2 -0.75 1.04 2.00 3.00 3.50 4.00 4.50 5.03 6.00 7.00 7.50 | 8.00 | 8.50 | 9.00 |
| 1 -0.74 1.00 2.00 3.00 3.50 4.00 4.49 5.00 6.00 7.00 7.50 | 8.00 | 8.50 | 9.00 |
| 2 -0.74 1.01 2.00 3.01 3.52 4.00 4.50 5.00 6.00 7.02 7.50 | 8.00 | 8.51 | 9.01 |
| 2 -0.74 1.01 2.00 3.00 3.51 4.00 4.50 5.00 6.00 7.01 7.51 | 8.00 | 8.50 | 9.01 |
| 3 -0.75 1.01 2.15 3.01 3.50 4.17 4.49 5.00 6.00 7.01 7.57 | 8.19 | 8.51 | 9.00 |
| 3 -0.75 1.00 2.01 3.00 3.50 4.00 4.51 5.00 6.00 7.01 7.52 | 8.01 | 8.50 | 9.00 |
| 1 -0.74 1.00 2.00 3.00 3.52 4.01 4.55 5.00 6.00 7.00 7.50 | 8.02 | 8.51 | 9.02 |
| 1 -0.75 1.00 2.00 3.00 3.55 4.01 4.50 5.00 6.00 7.00 7.50 | 8.02 | 8.52 | 9.01 |
| 2 -0.72 1.01 2.01 3.01 3.50 4.00 4.51 5.00 6.00 7.01 7.51 | 8.00 | 8.51 | 9.01 |
| 2 -0.72 1.01 2.00 3.01 3.50 4.00 4.50 5.00 6.00 7.00 7.50 | 8.00 | 8.51 | 9.02 |
| 1 -0.75 1.00 2.00 3.00 3.51 4.00 4.50 5.00 6.00 7.00 7.50 | 8.01 | 8.51 | 9.00 |
| 3 -0.75 1.00 2.00 3.00 3.50 4.00 4.50 5.00 6.00 7.00 7.52 | 8.01 | 8.52 | 9.02 |
| 3 -0.75 1.00 2.00 3.00 3.50 4.00 4.50 5.00 6.00 7.00 7.51 | 8.01 | 8.52 | 9.02 |

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix IV
Individual Subject Blood Sampling Times
Treatment B - EC Tablet Fed

| | | | | | | | Sc | cheduled | Time (h | ) ——— | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 9.5 | 10 | 12 | 14 | 16 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | 192 |
| PPD | | | | | | | | | | | | | | | |
| PPD | 1 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 1 | 9.51 | 10.00 | 12.00 | 14.00 | 16.00 | 24.06 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.01 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.01 | 72.00 | 96.21 | 120.09 | 144.01 | 168.09 | 192.00 |
| | 3 | 9.51 | 10.01 | 12.08 | 14.00 | 16.00 | 24.00 | 36.00 | 48.01 | 72.01 | 96.00 | 120.01 | 144.01 | 168.00 | 192.01 |
| | 3 | 9.50 | 10.01 | 12.02 | 14.00 | 16.00 | 24.00 | 36.05 | 48.00 | 72.01 | 96.00 | 120.01 | 144.01 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.00 | 12.00 | 14.01 | 16.02 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.07 | 144.00 | 168.02 | 192.01 |
| | 1 | 9.51 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.00 | 12.00 | 14.01 | 16.00 | 24.00 | 36.02 | 48.00 | 72.01 | 96.00 | 120.08 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.01 | 12.00 | 14.00 | 16.01 | 24.00 | 36.02 | 48.00 | 72.01 | 96.00 | 120.08 | 144.00 | 168.00 | 192.00 |
| | 3 | 9.50 | 10.01 | 12.00 | 14.13 | 16.00 | 24.00 | 36.06 | 48.00 | 72.01 | 96.24 | 120.01 | 144.00 | 168.00 | 192.00 |
| | 3 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.01 | 36.01 | 48.00 | 72.01 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 1 | 9.54 | 10.06 | 12.00 | 14.02 | 16.02 | 24.01 | 36.04 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.31 | 192.00 |
| | 1 | 9.54 | 10.00 | 12.00 | 14.02 | 16.01 | 24.00 | 36.01 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.51 | 10.01 | 12.01 | 14.01 | 16.00 | 24.01 | 36.03 | 48.00 | 72.01 | 96.02 | 120.09 | 144.00 | 168.01 | 192.03 |
| | 2 | 9.51 | 10.01 | 12.05 | 14.01 | 16.00 | 24.01 | 36.02 | 48.00 | 72.01 | 96.02 | 120.09 | 144.00 | 168.01 | 192.03 |
| | 1 | 9.54 | 10.00 | 12.00 | 14.02 | 16.02 | 24.00 | 36.08 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.02 | 192.01 |
| | 3 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.01 | 36.03 | 48.00 | 72.01 | 96.00 | 120.00 | 144.00 | 168.00 | 192.02 |
| | 3 | 9.50 | 10.00 | 12.01 | 14.00 | 16.00 | 24.00 | 36.10 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.01 |

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix IV
Individual Subject Blood Sampling Times
Treatment C - Uncoated Capsule + PPI Fasted

| | | | | | | | S | cheduled | Time (h) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 0 | 1 | 2 | 3 | 3.5 | 4 | 4.5 | 5 | 6 | 7 | 7.5 | 8 | 8.5 | 9 |
| PPD | | | | | | | | | | | | | | | |
| | 2 | -0.76 | 0.99 | 1.99 | 2.99 | 3.49 | 3.99 | 4.49 | 4.99 | 5.99 | 6.99 | 7.49 | 7.99 | 8.49 | 8.99 |
| | 3 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 3 | -0.64 | 1.06 | 2.06 | 3.08 | 3.55 | 4.01 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.70 | 9.00 |
| | 1 | -0.74 | 1.00 | 2.00 | 3.00 | 3.50 | 4.01 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 2 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.04 | 7.50 | 8.00 | 8.50 | 9.01 |
| | 1 | -0.77 | 1.00 | 2.02 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 2 | -0.75 | 1.00 | 2.00 | 3.00 | 3.55 | 4.00 | 4.50 | 5.00 | 6.00 | 7.02 | 7.56 | 8.00 | 8.50 | 9.02 |
| | 3 | -0.75 | 1.00 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.00 |
| | 1 | -0.75 | 1.00 | 2.00 | 3.00 | 3.51 | 4.14 | 4.51 | 5.00 | 6.00 | 7.00 | 7.50 | 8.15 | 8.50 | 9.00 |
| | 1 | -0.66 | 1.04 | 2.05 | 3.11 | 3.57 | 4.09 | 4.52 | 5.15 | 6.00 | 7.04 | 7.50 | 8.01 | 8.51 | 9.01 |
| | 2 | -0.73 | 1.01 | 2.01 | 3.01 | 3.52 | 4.00 | 4.51 | 5.00 | 6.00 | 7.01 | 7.51 | 8.02 | 8.51 | 9.00 |
| | 3 | -0.75 | 1.00 | 2.01 | 3.00 | 3.50 | 4.01 | 4.51 | 5.00 | 6.00 | 7.01 | 7.51 | 8.19 | 8.53 | 9.03 |
| | 3 | -0.75 | 1.00 | 2.01 | 3.04 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.01 | 7.54 | 8.01 | 8.51 | 9.01 |
| | 1 | -0.75 | 1.01 | 2.00 | 3.00 | 3.52 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.02 | 8.51 | 9.01 |
| | 3 | -0.75 | 1.00 | 2.01 | 3.00 | 3.50 | 4.01 | 4.50 | 5.00 | 6.00 | 7.00 | 7.52 | 8.01 | 8.55 | 9.02 |
| | 2 | -0.72 | 1.01 | 2.00 | 3.01 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.02 |
| | 1 | -0.75 | 1.00 | 2.00 | 3.00 | 3.51 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.01 | 8.51 | 9.00 |
| | 2 | -0.72 | 1.03 | 2.00 | 3.00 | 3.50 | 4.00 | 4.50 | 5.00 | 6.00 | 7.00 | 7.50 | 8.00 | 8.50 | 9.01 |

Wilson Therapeutics USA, Inc.
Study WTX101-102
July 14, 2014

Appendix IV
Individual Subject Blood Sampling Times
Treatment C - Uncoated Capsule + PPI Fasted

| | | | | | | | Sc | cheduled | Time (h | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | 9.5 | 10 | 12 | 14 | 16 | 24 | 36 | 48 | 72 | 96 | 120 | 144 | 168 | 192 |
| PPD | | | | | | | | | | | | | | | |
| PPD | 3 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.00 | 12.14 | 14.00 | 16.00 | 24.01 | 36.00 | 48.06 | 72.00 | 96.00 | 120.09 | 144.00 | 168.00 | 192.00 |
| | 1 | 9.52 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.01 | 48.00 | 72.01 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.01 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.01 | 72.00 | 96.01 | 120.09 | 144.01 | 168.01 | 192.01 |
| | 1 | 9.52 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.02 | 48.07 | 72.00 | 96.00 | 120.00 | 144.00 | 168.01 | 192.00 |
| | 3 | 9.50 | 10.00 | 12.00 | 14.05 | 16.00 | 24.00 | 36.05 | 48.00 | 72.00 | 96.00 | 120.01 | 144.00 | 168.00 | 192.00 |
| | 3 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 1 | 9.52 | 10.00 | 12.00 | 14.00 | 16.00 | 24.00 | 36.03 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 3 | 9.50 | 10.00 | 12.01 | 14.00 | 16.00 | 24.00 | 36.00 | 48.00 | 72.00 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.50 | 10.01 | 12.01 | 14.01 | 16.01 | 24.05 | 36.07 | 48.11 | 72.03 | 96.07 | 120.09 | 144.00 | 168.08 | 192.51 |
| | 1 | 9.53 | 10.01 | 12.00 | 14.02 | 16.03 | 24.01 | 36.06 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.01 | 192.00 |
| | 2 | 9.50 | 10.00 | 12.02 | 14.01 | 16.00 | 24.01 | 36.02 | 48.01 | 72.01 | 96.02 | 120.09 | 144.00 | 168.01 | 192.03 |
| | 2 | 9.51 | 10.03 | 12.03 | 14.01 | 16.00 | 24.01 | 36.01 | 48.01 | 72.01 | 96.02 | 120.09 | 144.00 | 168.01 | 192.03 |
| | 3 | 9.50 | 10.01 | 12.00 | 14.00 | 16.01 | 24.02 | 36.08 | 48.00 | 72.01 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 1 | 9.53 | 10.01 | 12.00 | 14.02 | 16.02 | 24.00 | 36.00 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.01 | 192.01 |
| | 3 | 9.50 | 10.00 | 12.00 | 14.00 | 16.00 | 24.01 | 36.10 | 48.00 | 72.01 | 96.00 | 120.00 | 144.00 | 168.00 | 192.00 |
| | 2 | 9.51 | 10.01 | 12.15 | 14.01 | 16.00 | 24.04 | 36.02 | 48.03 | 72.01 | 96.02 | 120.10 | 144.00 | 168.01 | 192.03 |
| | 1 | 9.53 | 10.00 | 12.00 | 14.02 | 16.01 | 24.00 | 36.10 | 48.01 | 72.00 | 96.00 | 120.00 | 144.00 | 168.03 | 192.00 |

 $\label{eq:power_power} \mbox{Appendix V}$  Descriptive Statistics for Plasma Concentrations

| | Schedule<br>Time | d · | A | rithmetic -<br>Standard | | Geome | tric | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | (h) | N | Mean | Error | CV (%) | Mean | CV (%) | Minimum | Median | Maximum |
| EC Tablet Fasted | 0.0 | 18 | 0.00 | 0.00 | | | | 0.00 | 0.00 | 0.00 |
| | 1.0 | 18 | 81.86 | 15.05 | 77.98 | 92.35 | 60.53 | 0.00 | 91.66 | 216.94 |
| | 2.0 | 18 | 182.41 | 19.36 | 45.02 | 175.93 | 53.28 | 0.00 | 201.62 | 291.58 |
| | 3.0 | 18 | 270.36 | 24.09 | 37.80 | 245.17 | 54.51 | 56.51 | 300.58 | 441.89 |
| | 3.5 | 18 | 299.14 | 26.82 | 38.04 | 270.50 | 55.52 | 62.06 | 309.38 | 429.67 |
| | 4.0 | 18 | 310.54 | 25.40 | 34.70 | 289.36 | 42.88 | 121.48 | 324.55 | 478.14 |
| | 4.5 | 18 | 342.70 | 24.25 | 30.02 | 326.06 | 35.03 | 147.29 | 356.11 | 533.87 |
| | 5.0 | 18 | 324.28 | 21.12 | 27.63 | 311.24 | 31.41 | 144.71 | 328.52 | 483.43 |
| | 6.0 | 18 | 330.35 | 21.16 | 27.17 | 316.70 | 32.59 | 127.97 | 339.31 | 483.92 |
| | 7.0 | 18 | 324.84 | 21.88 | 28.57 | 309.69 | 35.06 | 115.04 | 341.47 | 466.89 |
| | 7.5 | 18 | 324.69 | 21.45 | 28.03 | 310.16 | 34.26 | 116.83 | 332.96 | 471.67 |
| | 8.0 | 18 | 325.89 | 22.05 | 28.70 | 310.12 | 36.04 | 112.36 | 334.34 | 464.76 |
| | 8.5 | 18 | 318.34 | 20.98 | 27.96 | 304.37 | 33.76 | 117.64 | 326.48 | 484.69 |
| | 9.0 | 18 | 319.63 | 20.53 | 27.25 | 304.95 | 35.54 | 105.05 | 336.89 | 467.48 |
| | 9.5 | 18 | 329.17 | 22.02 | 28.39 | 313.74 | 35.40 | 112.76 | 344.61 | 483.93 |
| | 10.0 | 18 | 307.40 | 20.74 | 28.62 | 292.17 | 36.87 | 99.92 | 320.91 | 445.84 |
| | 12.0 | 18 | 289.40 | 20.69 | 30.33 | 273.61 | 38.60 | 95.51 | 307.20 | 441.49 |
| | 14.0 | 18 | 264.88 | 19.12 | 30.63 | 250.19 | 38.89 | 88.90 | 270.97 | 397.88 |
| | 16.0 | 18 | 247.80 | 18.48 | 31.63 | 232.93 | 40.76 | 79.60 | 264.01 | 371.79 |
| | 24.0 | 18 | 189.73 | 14.98 | 33.50 | 176.90 | 43.65 | 60.92 | 205.11 | 294.46 |
| | 36.0 | 18 | 144.48 | 11.63 | 34.15 | 133.98 | 45.73 | 47.59 | 156.72 | 217.24 |
| | 48.0 | 18 | 114.28 | 10.06 | 37.35 | 104.37 | 50.83 | 35.30 | 122.84 | 177.90 |
| | 72.0 | 18 | 74.04 | 7.16 | 41.04 | 66.50 | 55.59 | 21.94 | 78.14 | 115.16 |
| | 96.0 | 18 | 50.30 | 4.99 | 42.13 | 44.85 | 57.95 | 14.71 | 53.29 | 82.92 |
| | 120.0 | 18 | 36.09 | 3.58 | 42.07 | 32.33 | 56.16 | 10.78 | 37.58 | 65.42 |
| | 144.0 | 18 | 25.09 | 3.03 | 51.17 | 26.48 | 40.61 | 0.00 | 27.74 | 48.90 |
| | 168.0 | 18 | 18.54 | 2.41 | 55.12 | 21.44 | 28.93 | 0.00 | 21.13 | 36.43 |
| | 192.0 | 18 | 14.04 | 2.07 | 62.67 | 17.50 | 25.95 | 0.00 | 15.23 | 29.78 |

Geometric mean and CV were not calculated if all values were <LOQ Subject  $\stackrel{\mathsf{PPD}}{\mathsf{PPD}}$  Period 2, EC Tablet Fed, had a C(0) >= LOQ and >= 5% of Cmax and is excluded from the descriptive statistics.

 $\label{eq:power_power} \mbox{ Appendix V } \\ \mbox{ Descriptive Statistics for Plasma Concentrations } \\$ 

| | Schedule<br>Time | d - | A | rithmetic -<br>Standard | | Geome | tric | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | (h) | N | Mean | Error | CV (%) | Mean | CV (%) | Minimum | Median | Maximum |
| EC Tablet Fed | 0.0 | 17 | 0.00 | 0.00 | | | | 0.00 | 0.00 | 0.00 |
| | 1.0 | 17 | 33.39 | 9.69 | 119.66 | 38.03 | 105.08 | 0.00 | 17.63 | 122.88 |
| | 2.0 | 17 | 80.25 | 18.74 | 96.30 | 76.30 | 119.59 | 0.00 | 62.27 | 223.00 |
| | 3.0 | 17 | 121.06 | 24.10 | 82.07 | 104.20 | 101.13 | 0.00 | 81.62 | 295.07 |
| | 3.5 | 17 | 144.02 | 27.38 | 78.39 | 125.02 | 101.16 | 0.00 | 103.86 | 338.70 |
| | 4.0 | 17 | 150.94 | 28.60 | 78.13 | 132.02 | 97.60 | 0.00 | 122.75 | 365.88 |
| | 4.5 | 17 | 161.07 | 29.70 | 76.01 | 144.91 | 88.26 | 0.00 | 137.05 | 386.35 |
| | 5.0 | 17 | 157.43 | 27.02 | 70.76 | 113.75 | 117.40 | 12.85 | 130.62 | 369.95 |
| | 6.0 | 17 | 161.16 | 25.06 | 64.12 | 125.81 | 93.17 | 21.31 | 136.16 | 362.28 |
| | 7.0 | 17 | 163.23 | 24.69 | 62.38 | 129.52 | 87.59 | 26.61 | 125.60 | 355.71 |
| | 7.5 | 17 | 160.05 | 24.60 | 63.37 | 127.12 | 86.46 | 27.15 | 124.38 | 357.16 |
| | 8.0 | 17 | 158.82 | 25.02 | 64.95 | 124.80 | 88.86 | 26.70 | 121.14 | 362.04 |
| | 8.5 | 17 | 151.68 | 23.78 | 64.65 | 119.71 | 87.91 | 24.40 | 112.86 | 351.14 |
| | 9.0 | 17 | 150.80 | 24.12 | 65.95 | 118.01 | 89.98 | 23.84 | 118.34 | 361.03 |
| | 9.5 | 17 | 149.23 | 24.67 | 68.16 | 115.88 | 91.40 | 22.74 | 119.70 | 387.75 |
| | 10.0 | 17 | 137.83 | 22.91 | 68.53 | 106.54 | 92.83 | 20.35 | 112.78 | 361.80 |
| | 12.0 | 17 | 123.76 | 21.65 | 72.13 | 92.96 | 100.39 | 15.83 | 104.55 | 336.48 |
| | 14.0 | 17 | 109.98 | 19.25 | 72.15 | 81.35 | 105.94 | 12.49 | 95.49 | 287.92 |
| | 16.0 | 17 | 95.94 | 17.72 | 76.18 | 79.68 | 86.97 | 0.00 | 83.22 | 271.27 |
| | 24.0 | 17 | 70.46 | 13.43 | 78.60 | 57.43 | 91.87 | 0.00 | 59.42 | 205.55 |
| | 36.0 | 17 | 50.22 | 10.52 | 86.33 | 39.03 | 102.04 | 0.00 | 36.81 | 164.40 |
| | 48.0 | 17 | 38.07 | 8.02 | 86.84 | 33.62 | 85.70 | 0.00 | 28.19 | 123.25 |
| | 72.0 | 17 | 23.88 | 5.35 | 92.33 | 26.27 | 66.86 | 0.00 | 17.43 | 81.51 |
| | 96.0 | 17 | 15.08 | 3.47 | 94.78 | 21.20 | 48.34 | 0.00 | 12.95 | 46.99 |
| | 120.0 | 17 | 10.86 | 2.60 | 98.70 | 17.34 | 38.81 | 0.00 | 11.03 | 31.11 |
| | 144.0 | 17 | 6.52 | 2.06 | 130.16 | 15.31 | 28.41 | 0.00 | 0.00 | 22.42 |
| | 168.0 | 17 | 4.75 | 1.64 | 142.69 | 13.25 | 19.31 | 0.00 | 0.00 | 16.87 |
| | 192.0 | 17 | 3.08 | 1.40 | 187.00 | 13.05 | 11.52 | 0.00 | 0.00 | 14.61 |

Geometric mean and CV were not calculated if all values were <LOQ Subject  $\stackrel{\mathsf{PPD}}{\mathsf{PPD}}$  Period 2, EC Tablet Fed, had a C(0) >= LOQ and >= 5% of Cmax and is excluded from the descriptive statistics.

 $\label{eq:power_power} \mbox{Appendix V}$  Descriptive Statistics for Plasma Concentrations

| | Scheduled - Time | | | | —<br>—— Geometric —— | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | (h) | N | Mean | Error | CV (%) | Mean | CV (%) | Minimum | Median | Maximum |
| | 0.0 | 1.0 | 0.55 | 0.55 | 404.06 | 10.00 | | 0.00 | 0.00 | 10.00 |
| Uncoated Capsule + PPI Fasted | 0.0 | 18 | 0.57 | 0.57 | 424.26 | 10.28 | 01 01 | 0.00 | 0.00 | 10.28 |
| | 1.0 | 18 | 207.87 | 10.32 | 21.07 | 203.45 | 21.81 | 127.23 | 203.70 | 292.36 |
| | 2.0 | 18<br>18 | 302.26 | 12.64 | 17.74 | 297.80 | 17.91 | 226.09 | 302.76 | 414.18 |
| | 3.0<br>3.5 | 18 | 372.60<br>390.04 | 14.83 | 16.88<br>15.92 | 367.45<br>385.41 | 17.47<br>16.02 | 261.60<br>281.36 | 373.18<br>383.33 | 496.93<br>525.94 |
| | 4.0 | | | 14.64 | | | | | | 514.24 |
| | 4.0 | 18<br>18 | 400.26<br>424.85 | 15.18 | 16.09 | 395.34 | 16.37<br>17.33 | 286.07 | 401.09 | 567.10 |
| | | | | 17.35 | 17.33 | 418.94 | | 313.14 | 420.93 | |
| | 5.0 | 18 | 395.88 | 15.74 | 16.87 | 390.66 | 16.86 | 285.64 | 390.05 | 522.42 |
| | 6.0 | 18 | 384.51 | 13.92 | 15.36 | 380.26 | 15.47 | 278.19 | 386.99 | 500.18 |
| | 7.0 | 18 | 377.58 | 12.56 | 14.11 | 374.05 | 14.22 | 281.49 | 377.80 | 484.56 |
| | 7.5 | 18 | 375.58 | 13.13 | 14.83 | 371.75 | 14.79 | 291.78 | 377.98 | 490.01 |
| | 8.0 | 18 | 372.67 | 11.39 | 12.97 | 369.69 | 13.17 | 296.67 | 371.46 | 457.84 |
| | 8.5 | 18 | 378.41 | 12.10 | 13.56 | 375.07 | 13.87 | 288.49 | 384.04 | 466.42 |
| | 9.0 | 18 | 373.10 | 12.47 | 14.18 | 369.52 | 14.44 | 283.64 | 375.52 | 469.08 |
| | 9.5 | 18 | 381.32 | 12.45 | 13.85 | 377.85 | 14.03 | 289.70 | 377.79 | 479.68 |
| | 10.0 | 18 | 363.25 | 13.36 | 15.60 | 359.02 | 15.96 | 273.28 | 362.16 | 475.05 |
| | 12.0 | 18 | 343.08 | 13.11 | 16.21 | 338.90 | 16.23 | 251.68 | 346.36 | 483.18 |
| | 14.0 | 18 | 314.88 | 13.45 | 18.12 | 310.20 | 17.85 | 227.71 | 309.92 | 444.36 |
| | 16.0 | 18 | 292.20 | 11.95 | 17.35 | 288.16 | 17.26 | 210.72 | 290.22 | 411.71 |
| | 24.0 | 18 | 229.57 | 10.04 | 18.55 | 225.89 | 18.70 | 158.07 | 226.98 | 331.55 |
| | 36.0 | 18 | 177.41 | 7.05 | 16.86 | 175.04 | 17.05 | 128.40 | 179.96 | 248.04 |
| | 48.0 | 18 | 138.97 | 5.88 | 17.96 | 136.86 | 18.21 | 95.76 | 137.02 | 191.50 |
| | 72.0 | 18 | 92.13 | 4.55 | 20.97 | 90.18 | 21.81 | 56.85 | 88.74 | 125.29 |
| | 96.0 | 18 | 61.54 | 3.65 | 25.17 | 59.66 | 26.41 | 35.40 | 59.59 | 86.90 |
| | 120.0 | 18 | 42.91 | 2.63 | 25.98 | 41.57 | 26.56 | 24.03 | 42.01 | 66.86 |
| | 144.0 | 18 | 34.59 | 3.69 | 45.29 | 32.00 | 40.74 | 16.75 | 31.53 | 84.79 |
| | 168.0 | 18 | 24.17 | 1.75 | 30.79 | 23.08 | 32.43 | 12.92 | 22.81 | 36.86 |
| | 192.0 | 18 | 18.14 | 1.33 | 31.18 | 17.33 | 31.86 | 10.21 | 17.48 | 28.30 |

Geometric mean and CV were not calculated if all values were <LOQ Subject  $\stackrel{\mathsf{PPD}}{\mathsf{PPD}}$  Period 2, EC Tablet Fed, had a C(0) >= LOQ and >= 5% of Cmax and is excluded from the descriptive statistics.

Appendix VI
Individual Subject Pharmacokinetic Parameters
Treatment A - EC Tablet Fasted

| Subject | Period | Lag<br>Time*<br>(h) | CMAX<br>(ng/mL) | TMAX<br>(h) | AUC(0-t)<br>(hxng/mL) | AUC(inf)<br>(hxng/mL) | % AUC<br>Extrap | Regre<br>Start<br>Nominal | Time | Final<br>Time<br>C>=LOQ | No. Points<br>in Regr | Regr<br>r² | Lambda_z | t½<br>(h) | CL/F<br>(L/h) | Vz/F<br>(L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | | | | | | | | | | | | | | | | |
| | 3 | • | 147.29 | | 4,857.67 | | | 47.00 | 48.00 | 120.00 | | | 0.01649 | | 2.415 | 146.42 |
| | 2 | • | 269.11 | | 11,565.25 | , | | 71.00 | 72.00 | 168.00 | | | 0.01444 | | 1.068 | 74.02 |
| | 1 | • | 278.51 | | 7,607.44 | , | | 47.00 | 48.00 | 120.00 | 4 | | 0.01954 | | 1.611 | 82.45 |
| | 2 | • | 441.89 | | 16,120.60 | , | | 47.00 | 48.01 | 192.01 | 7 | | 0.01418 | | 0.775 | 54.66 |
| | 1 | 3.00 | 397.87 | | 18,547.33 | , | | 48.00 | 48.07 | 192.00 | | | 0.01406 | | 0.672 | 47.77 |
| | 3 | | 450.27 | | 22,675.96 | , | | 36.00 | 36.05 | 192.00 | | | 0.01175 | | 0.528 | 44.91 |
| | 3 | | 483.93 | | 22,738.24 | , | | 36.00 | 36.00 | 192.00 | | | 0.01476 | | 0.550 | 37.29 |
| | 1 | | 411.20 | 3.52 | 19,268.61 | 20,226.41 | 4.7 | 23.00 | 24.00 | 192.00 | 9 | 0.9983 | 0.01587 | 43.69 | 0.658 | 41.47 |
| | 3 | 2.00 | 450.94 | 6.00 | 18,755.35 | 19,781.67 | 5.2 | 72.00 | 72.00 | 192.00 | 6 | 0.9926 | 0.01456 | 47.62 | 0.673 | 46.22 |
| | 2 | | 424.72 | 4.55 | 16,498.83 | 18,491.08 | 10.8 | 96.00 | 96.07 | 192.51 | 5 | 0.9952 | 0.00974 | 71.13 | 0.720 | 73.86 |
| | 1 | | 382.79 | 9.53 | 19,676.87 | 21,468.36 | 8.3 | 36.00 | 36.06 | 192.00 | 8 | 0.9879 | 0.01315 | 52.69 | 0.620 | 47.13 |
| | 2 | | 445.60 | 4.53 | 18,779.74 | 19,761.83 | 5.0 | 36.00 | 36.02 | 192.03 | 8 | 0.9910 | 0.01573 | 44.07 | 0.673 | 42.82 |
| | 2 | | 370.37 | 9.51 | 19,630.94 | 20,973.13 | 6.4 | 36.00 | 36.01 | 192.03 | 8 | 0.9896 | 0.01441 | 48.09 | 0.635 | 44.02 |
| | 3 | | 392.60 | 4.00 | 14,002.34 | 15,276.58 | 8.3 | 95.00 | 96.00 | 192.00 | 5 | 0.9508 | 0.01078 | 64.31 | 0.871 | 80.83 |
| | 1 | | 355.54 | 6.00 | 11,500.16 | 12,493.18 | 7.9 | 95.00 | 96.00 | 192.01 | 5 | 0.9979 | 0.01105 | 62.72 | 1.065 | 96.40 |
| | 3 | 2.00 | 219.93 | 7.52 | 6,732.08 | 7,574.44 | 11.1 | 72.00 | 72.01 | 144.00 | 4 | 0.9866 | 0.01201 | 57.70 | 1.757 | 146.27 |
| | 2 | | 312.57 | 4.50 | 15,414.33 | 16,514.39 | 6.7 | 36.00 | 36.02 | 192.03 | 8 | 0.9886 | 0.01387 | 49.98 | 0.806 | 58.11 |
| | 1 | 2.00 | 533.87 | | 24,102.97 | , | | 36.00 | 36.10 | 192.00 | | 0.9947 | 0.01522 | | 0.522 | 34.31 |

<sup>(. =</sup> parameter could not be estimated)

<sup>\*</sup>A lag time was not calculated if the first concentration >= LOQ occurred at the first sample time.

Appendix VI Individual Subject Pharmacokinetic Parameters Treatment B - EC Tablet Fed

| Subject | t Period | Lag<br>Time*<br>(h) | CMAX<br>(ng/mL) | TMAX<br>(h) | AUC(0-t) (hxng/mL) | AUC(inf)<br>(hxng/mL) | % AUC<br>Extrap | Regres<br>Start<br>Nominal | Time | Final<br>Time<br>C>=LOQ | No. Points<br>in Regr | Regr<br>r² | Lambda_z<br>(/h) | t½<br>(h) | CL/F<br>(L/h) | Vz/F<br>(L) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| PPD | | - 00 | 07.15 | | 100.00 | 070.10 | 24.5 | 0.00 | 0.50 | 14.00 | | | 0 10001 | | 47.60 | 267 22 |
| | 1 | 5.00 | 27.15 | 7.50 | | | | 9.00 | 9.50 | 14.00 | | | 0.12981 | | 47.68 | 367.33 |
| | 1 | 2.00 | 144.33 | 4.50 | | 3,402.37 | | 35.00 | 36.00 | 72.00 | | | 0.02326 | | 3.912 | 168.16 |
| | 2 | 3.00 | 71.48 | | 1,399.14 | , | | 16.00 | 16.00 | 48.01 | 4 | | 0.03703 | | 7.738 | 208.96 |
| | 3 | • | 387.75 | | 17,013.40 | , | 5.4 | 72.00 | 72.01 | 192.01 | 6 | 0.9690 | 0.01449 | 47.83 | 0.740 | 51.06 |
| | 3 | | 75.27 | 7.00 | 1,609.92 | | | | | 72.01 | | | | | | |
| | 2 | | 30.39 | 8.00 | 2,549.77 | 4,919.52 | 48.2 | 35.00 | 36.00 | 168.02 | 7 | 0.9893 | 0.00433 | 160.09 | 2.705 | 624.84 |
| | 1 | | 45.72 | 7.00 | 763.11 | 1,018.73 | 25.1 | 15.00 | 16.00 | 36.00 | 3 | 0.9875 | 0.03948 | 17.56 | 13.06 | 330.94 |
| | 2 | | 278.69 | 3.52 | 7,424.04 | 8,387.45 | 11.5 | 47.00 | 48.00 | 168.00 | 6 | 0.9627 | 0.01195 | 57.98 | 1.587 | 132.74 |
| | 2 | 5.00 | 315.30 | 8.00 | 11,538.14 | 12,881.72 | 10.4 | 72.00 | 72.01 | 192.00 | 6 | 0.9511 | 0.01087 | 63.75 | 1.033 | 95.02 |
| | 3 | 2.15 | 250.60 | 7.01 | 8,727.92 | 9,907.93 | 11.9 | 72.00 | 72.01 | 192.00 | 6 | 0.9625 | 0.00970 | 71.44 | 1.343 | 138.45 |
| | 3 | | 73.25 | 6.00 | 2,726.49 | | | | | 120.00 | | | | | | |
| | 1 | 3.00 | 314.87 | 4.55 | | 10,528.76 | | 48.00 | 48.01 | 168.31 | 6 | 0.9841 | 0.01609 | 43.08 | 1.264 | 78.56 |
| | 1 | | 256.51 | 4.50 | | 7,909.66 | | 48.00 | 48.01 | 144.00 | 5 | 0.9857 | 0.01477 | 46.92 | 1.683 | 113.89 |
| | 2 | | 137.05 | 4.51 | | , | | 36.00 | 36.03 | 96.02 | | | 0.01752 | | 2.693 | 153.70 |
| | 2 | | 87.43 | 4.50 | | , | | 24.00 | 24.01 | 48.00 | | | 0.02677 | | 6.342 | 236.93 |
| | 1 | • | 272.07 | 4.50 | • | , | | 48.00 | 48.01 | 120.00 | | | 0.01567 | | 1.762 | 112.43 |
| | 3 | • | 108.85 | | 3,163.41 | , | | 48.00 | 48.00 | 120.00 | | | 0.01367 | | 3.129 | 324.50 |
| | 3 | • | | | | , | | | | | | | | | | |
| | 3 | | 325.45 | 4.50 | 10,511.03 | 11,/30.88 | 10.4 | 72.00 | 72.00 | 192.01 | 6 | 0.9850 | 0.01007 | 68.83 | 1.135 | 112.66 |

<sup>(. =</sup> parameter could not be estimated)

<sup>\*</sup>A lag time was not calculated if the first concentration >= LOQ occurred at the first sample time.

Appendix VI Individual Subject Pharmacokinetic Parameters Treatment C - Uncoated Capsule + PPI Fasted

| | | Lag | | | | | | Regre | ssion | Final | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Period | Time* (h) | CMAX<br>(ng/mL) | TMAX<br>(h) | AUC(0-t)<br>(hxng/mL) | AUC(inf)<br>(hxng/mL) | % AUC<br>Extrap | Start<br>Nominal | | Time<br>C>=LOQ | No. Points<br>in Regr | Regr<br>r² | Lambda_z<br>(/h) | t½<br>(h) | CL/F<br>(L/h) | Vz/F<br>(L) |
| PPD | | | | | | | | | | | | | | | | |
| | 2 | | 445.77 | 2.99 | 20,896.85 | • | | • | • | 191.99 | | - | | | | • |
| | 3 | | 353.87 | 3.50 | 13,764.48 | 14,481.24 | 4.9 | 72.00 | 72.00 | 192.00 | 6 | 0.9832 | 0.01425 | 48.65 | 0.919 | 64.50 |
| | 3 | | 447.08 | 4.50 | 16,092.90 | 16,804.88 | 4.2 | 48.00 | 48.00 | 192.10 | 7 | 0.9851 | 0.01599 | 43.36 | 0.792 | 49.54 |
| | 1 | | 460.34 | 4.50 | 17,746.68 | 18,479.64 | 4.0 | 35.00 | 36.00 | 192.00 | 8 | 0.9913 | 0.01683 | 41.18 | 0.720 | 42.78 |
| | 2 | | 420.63 | 10.01 | 24,901.94 | 27,095.86 | 8.1 | 36.00 | 36.03 | 192.01 | 8 | 0.9972 | 0.01290 | 53.74 | 0.491 | 38.08 |
| | 1 | | 402.97 | 4.50 | 22,358.35 | 24,570.85 | 9.0 | 36.00 | 36.00 | 192.01 | 8 | 0.9932 | 0.01236 | 56.07 | 0.542 | 43.81 |
| | 2 | | 459.34 | 4.50 | 19,914.87 | 21,093.09 | 5.6 | 35.00 | 36.00 | 192.00 | 8 | 0.9884 | 0.01490 | 46.51 | 0.631 | 42.34 |
| | 3 | | 367.72 | 4.50 | 15,920.08 | 16,873.34 | 5.6 | 36.00 | 36.04 | 192.00 | 8 | 0.9921 | 0.01484 | 46.71 | 0.789 | 53.16 |
| | 1 | | 477.57 | 3.51 | 21,464.59 | 22,684.16 | 5.4 | 23.00 | 24.00 | 192.00 | 9 | 0.9913 | 0.01519 | 45.64 | 0.587 | 38.63 |
| | 1 | | 566.16 | 4.52 | 27,087.62 | 29,032.66 | 6.7 | 36.00 | 36.15 | 192.08 | 8 | 0.9877 | 0.01402 | 49.43 | 0.458 | 32.69 |
| | 2 | | 375.17 | 5.00 | 19,190.70 | 20,783.64 | 7.7 | 36.00 | 36.02 | 192.01 | 8 | 0.9857 | 0.01316 | 52.69 | 0.640 | 48.68 |
| | 3 | | 496.93 | 3.00 | 18,655.05 | 19,475.16 | 4.2 | 24.00 | 24.00 | 192.00 | 9 | 0.9905 | 0.01656 | 41.85 | 0.683 | 41.26 |
| | 3 | | 405.34 | 4.00 | 20,677.13 | 22,327.76 | 7.4 | 24.00 | 24.00 | 192.00 | 9 | 0.9941 | 0.01382 | 50.15 | 0.596 | 43.13 |
| | 1 | | 567.10 | 4.50 | 19,428.23 | 20,907.70 | 7.1 | 95.00 | 96.00 | 192.01 | 5 | 0.9743 | 0.01177 | 58.91 | 0.637 | 54.10 |
| | 3 | | 406.89 | 9.02 | 18,674.17 | 19,730.51 | 5.4 | 24.00 | 24.01 | 192.00 | 9 | 0.9945 | 0.01514 | 45.78 | 0.675 | 44.55 |
| | 2 | | 525.94 | 3.50 | 23,040.95 | 24,447.55 | 5.8 | 36.00 | 36.04 | 192.03 | 8 | 0.9818 | 0.01495 | 46.37 | 0.544 | 36.42 |
| | 1 | | 313.14 | | 14,392.65 | , | | 23.00 | 24.00 | 192.00 | 9 | | 0.01531 | 45.28 | 0.872 | 56.94 |
| | 2 | | 460.65 | | 22,362.06 | , | | 24.00 | 24.00 | 192.03 | 9 | | 0.01490 | | 0.560 | 37.60 |

<sup>(. =</sup> parameter could not be estimated)

 $<sup>^{*}</sup>$ A lag time was not calculated if the first concentration >= LOQ occurred at the first sample time.

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix VII
Descriptive Statistics for Pharmacokinetic Parameters

| | | | | A1 | rithmetic — | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Standard | | Geometr | ic | | | |
| Treatment | Parameter | Units | N | Mean | Deviation | CV (%) | Mean | CV (%) | Minimum | Median | Maximum |
| DC Mahlat Dastad | TLAG | h | 4 | 2.2513 | 0 5010 | 22.26 | | | 1 0004 | 2 0014 | 3.0031 |
| EC Tablet Fasted | CMAX | na/mL | 4<br>18 | 376.0559 | 98.0308 | 22.26 | | 20 52 | | | |
| | TMAX | ng/шь<br>h | 18 | 5.8976 | 2.2000 | | | | | | |
| | | | | | | | | 47.45 | 3.0036 | | |
| | AUC(0-t) | | | | | | 14,790.8396 | | | | |
| | AUC(inf) | _ | | | | | 15,997.7562 | | | | |
| | Lambda_z | /h | 18 | 0.0140 | | 16.74 | | 17.10 | | | |
| | t½ | h<br>- '' | 18 | 50.9539 | | 17.41 | | | | | |
| | CL/F | L/h | 18 | 0.9233 | | | | | | | |
| | Vz/F | L | 18 | 66.6092 | 33.9633 | 50.99 | 60.3180 | 45.88 | 34.3132 | 51.2159 | 146.4164 |
| EC Tablet Fed | TLAG | h | 6 | 3.3586 | 1.3386 | 39.86 | • | | 1.9994 | 3.0015 | 5.0017 |
| | CMAX | ng/mL | 17 | 186.5738 | 117.6370 | 63.05 | 145.1312 | 94.12 | 27.1480 | 144.3250 | 387.7480 |
| | TMAX | h | 17 | 5.8001 | 1.6925 | 29.18 | | | 3.5161 | 4.5542 | 9.5056 |
| | AUC(0-t) | hxng/mL | 17 | 5,740.3997 | 4,680.9190 | 81.54 | 3,635.5289 | 170.21 | 182.9003 | 4,203.4749 | 17,013.3966 |
| | AUC(inf) | hxng/mL | 15 | 6,973.4432 | 5,065.3161 | 72.64 | 4,654.6700 | 160.02 | 279.1198 | 7,554.0780 | 17,986.4628 |
| | Lambda z | /h | 15 | 0.0258 | 0.0303 | 117.32 | 0.0189 | 79.66 | 0.0096 | 0.0157 | 0.1298 |
| | t½ | h | 15 | 43.5216 | 20.9345 | 48.10 | 36.7348 | 79.66 | 5.3398 | 44.2336 | 71.8877 |
| | CL/F | L/h | 15 | 6.3404 | 11.9177 | 187.96 | 2.8593 | 160.02 | 0.7399 | 1.7618 | 47.6820 |
| | Vz/F | L | 15 | 175.0215 | 98.1477 | 56.08 | 151.5334 | 60.81 | 51.0613 | 138.4459 | 367.3285 |
| Uncoated Capsule + PPI Fasted | TLAG | h | 0 | | | | | | | | |
| | CMAX | ng/mL | 18 | 441.8128 | 69.5915 | | | | | | |
| | TMAX | h . | 18 | 4.7257 | | 39.03 | | | 2.9919 | | |
| | AUC(0-t) | hxna/mT | 18 | 19.809.4048 | | | 19,511.1356 | 18.23 | | | |
| | AUC(inf) | | | | | | 20,682.9228 | | | | |
| | Lambda z | /h | 17 | • | 0.0014 | | , | | | , | • |
| | t½ | h | 17 | | | 10.10 | | | | | |
| | CL/F | L/h | 17 | 0.6551 | | 19.74 | | | | | |
| | Vz/F | L | 17 | 45.1889 | | 18.39 | | | | | |

Geometric mean and CV were not calculated for Tmax or Tlag. Subject  $\overline{PPD}$  Period 2, EC Tablet Fed, had a C(0) >= LOQ and >= 5% of Cmax and is excluded from the descriptive statistics.

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

## Appendix VIII Statistical Analysis of Pharmacokinetic Parameters

The GLM Procedure

Class Level Information

| Class | Levels | Values |
|-----------|---------|--------------------------------------------------|
| SUBJECT | 18 | PPD |
| PERIOD | 3 | 1 2 3 |
| TREATMENT | 3 | АВС |
| SEQUENCE | 6 | ABC ACB BAC BCA CAB CBA |
| | Data fo | or Analysis of LNCMAX LNAUCT |
| | | f Observations Read 53<br>f Observations Used 53 |
| | Da | ta for Analysis of LNAUC |

Number of Observations Read Number of Observations Used 53

50

NOTE: Variables in each group are consistent with respect to the presence or absence of missing values.

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

## Appendix VIII Statistical Analysis of Pharmacokinetic Parameters

The GLM Procedure

Dependent Variable: LNCMAX

| Source | DF | Sum of<br>Squares Mea | n Square F | Value | Pr > F |
|---|---|---|---|---|---|
| Model | 21 17. | 88490026 0. | 85166192 | 4.11 | 0.0002 |
| Error | 31 6. | 42240550 0. | 20717437 | | |
| Corrected Total | 52 24. | 30730576 | | | |
| R-Square | Coeff Var | Root MSE | LNCMAX Mean | | |
| 0.735783 | 8.040249 | 0.455164 | 5.661070 | | |
| Source | DF Typ | e III SS Mea | n Square F | Value | Pr > F |
| SEQUENCE<br>SUBJECT (SEQUENCE)<br>PERIOD<br>TREATMENT | 12 4.<br>2 0. | 05190490 0.<br>02154484 0. | | 1.63 | 0.1668<br>0.1341<br>0.9494<br><.0001 |
| Tests of Hypotheses Using | | | | | |
| Source<br>SEQUENCE | | e III SS Mea<br>74914402 0. | - | | Pr > F<br>0.4401 |
| Parameter | Estima | Standa<br>te Err | | Pr > | t |
| B-A<br>A-C | -0.904196<br>-0.190497 | 0.155236<br>75 0.151721 | | <.00<br>0.21 | |

Wilson Therapeutics USA, Inc.
Study WTX101-102
July 14, 2014

## Appendix VIII Statistical Analysis of Pharmacokinetic Parameters

The GLM Procedure

Dependent Variable: LNAUCT

| Source | DF | Sum o | | quare F | Value | Pr > F |
|---|---|---|---|---|---|---|
| Model | 21 | 40.442383 | 85 1.925 | 82780 | 4.43 | <.0001 |
| Error | 31 | 13.466791 | 28 0.434 | 41262 | | |
| Corrected Total | 52 | 53.909175 | 13 | | | |
| R-Squar | e Coef: | f Var 1 | Root MSE LI | NAUCT Mean | | |
| 0.75019 | 5 7.12 | 28694 | 0.659100 | 9.245731 | | |
| Source | DF | Type III : | SS Mean So | quare F | Value | Pr > F |
| SEQUENCE<br>SUBJECT (SEQUENCE)<br>PERIOD<br>TREATMENT | | 5.151345;<br>6.806517;<br>0.404451;<br>26.680463; | 09 0.5672<br>89 0.2022 | 22595 | 2.37<br>1.31<br>0.47<br>30.71 | 0.0621<br>0.2646<br>0.6321<br><.0001 |
| Tests of Hypotheses Us | - | | | | | |
| Source | DF | Type III : | | quare F | | Pr > F |
| SEQUENCE | 5 | 5.151345 | 33 1.030 | 26907 | 1.82 | 0.1840 |
| Parameter | Es | stimate | Standard<br>Error | t Value | Pr > | t |
| B-A<br>A-C | | 7848178<br>7697732 | 0.22479020<br>0.21969995 | | | |

# Appendix VIII Statistical Analysis of Pharmacokinetic Parameters

The GLM Procedure Least Squares Means

| TREATMENT | LNCMAX<br>LSMEAN |
|-------------|----------------------------------------|
| A<br>B<br>C | 5.88855268<br>4.98435657<br>6.07905043 |
| TREATMENT | LNAUCT<br>LSMEAN |
| A<br>B<br>C | 9.60176332<br>8.22328154<br>9.87874064 |

Wilson Therapeutics USA, Inc.
Study WTX101-102
July 14, 2014

## Appendix VIII Statistical Analysis of Pharmacokinetic Parameters

------ ASSAY=Total Molybdenum ------

The GLM Procedure

Dependent Variable: LNAUC

| Source | Sum<br>DF Squar | | F Value Pr > F |
|---|---|---|---|
| Model | 21 34.118775 | 40 1.62470359 | 6.09 <.0001 |
| Error | 28 7.470801 | 00 0.26681432 | |
| Corrected Total | 49 41.589576 | 41 | |
| R-Square | Coeff Var | Root MSE LNAUC Mean | ו |
| 0.820368 | 5.496773 | 0.516541 9.397163 | 3 |
| Source | DF Type III | SS Mean Square 1 | F Value Pr > F |
| SEQUENCE<br>SUBJECT (SEQUENCE)<br>PERIOD<br>TREATMENT | 5 7.442085<br>12 7.761184<br>2 0.593164<br>2 14.447876 | 63 0.64676539<br>63 0.29658231 | 5.58 0.0011<br>2.42 0.0263<br>1.11 0.3431<br>27.07 <.0001 |
| Tests of Hypotheses Using | the Type III MS f | or SUBJECT(SEQUENCE) as | an Error Term |
| Source | DF Type III | SS Mean Square I | F Value Pr > F |
| SEQUENCE | 5 7.442085 | 65 1.48841713 | 2.30 0.1100 |
| Parameter | Estimate | Standard<br>Error t Value | e Pr > t |
| B-A<br>A-C | -1.14888271<br>-0.13736930 | 0.18557883 -6.19<br>0.17620792 -0.79 | 9 <.0001<br>8 0.4422 |

## Appendix VIII Statistical Analysis of Pharmacokinetic Parameters

------ ASSAY=Total Molybdenum ------

The GLM Procedure Least Squares Means

| TREATMENT | LNAUC LSMEAN |
|-----------|--------------|
| A | 9.68020375 |
| В | 8.53132104 |
| C | 9.81757305 |

Wilson Therapeutics USA, Inc.

Study WTX101-102

July 14, 2014

Appendix VII
Statistical Analysis of Pharmacokinetic Parameters

| | - | Geometric Means | | - Geometric - 90% Confid | | Within<br>ence Interval — Subject Power* | | |
|---|---|---|---|---|---|---|---|---|
| Comparison | Parameter | Test | Reference | Mean Ratio | Lower Limit | Upper Limit | CV (%) | (%) |
| B-A | CMAX | 146.11 | 360.88 | 40.49 | 31.12 | 52.68 | 47.98 | 67.14 |
| | AUC(0-t) | 3,726.71 | 14,790.84 | 25.20 | 17.21 | 36.89 | 73.76 | 77.30 |
| | AUC(inf) | 5,071.14 | 15,997.76 | 31.70 | 23.12 | 43.47 | 55.30 | 72.58 |
| A-C | CMAX | 360.88 | 436.61 | 82.65 | 63.91 | 106.90 | 47.98 | 66.48 |
| | AUC(0-t) | 14,790.84 | 19,511.14 | 75.81 | 52.23 | 110.02 | 73.76 | 76.76 |
| | AUC(inf) | 15,997.76 | 18,353.45 | 87.16 | 64.59 | 117.63 | 55.30 | 71.10 |

Data were natural log-transformed before analysis. \*Power to detect a 20% difference at alpha = 0.05.

tment A - EC Tablet Fasted; Treatment B - EC Tablet Fed; Treatment C - Uncoated Capsule + PPI Fasted Subject  $\stackrel{\mathsf{PPD}}{\mathsf{PPD}}$  Period 2, EC Tablet Fed, had a C(0) >= LOQ and >= 5% of Cmax and is excluded from the statistical analyses.



Uncoated Capsule + PPI Fasted

Time (hr)

▲▲▲EC Tablet Fed

Uncoated Capsule + PPI Fasted

Time (hr)

AAA EC Tablet Fed













Time (hr)

Uncoated Capsule + PPI Fasted

▲▲▲EC Tablet Fed

100-

Uncoated Capsule + PPI Fasted

96

AAA EC Tablet Fed

Time (hr)





Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes


Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



Appendix X — Individual Subject Total Mo Concentration vs. Time Graphs — Semi-Logarithmic Axes



## 16.1.9.2 Statistical Methods

## 16.1.9.2.1 Statistical Analysis Plan

## **Statistical Analysis Plan**

A Phase 1, Single-Center, Randomized, 3-Period Crossover Study in Healthy Volunteers to Evaluate the Absorption of WTX101 After Single Dose Administration of an Enteric Coated Formulation with and without food and a Non-Coated Formulation Coadministered with a Proton Pump Inhibitor without Food

Protocol No. WTX101-102 Celerion Project CA13895

Final Version 1.0 Date: 12 May 2014

Compound Name: WTX101

Final Protocol Date: 25 February 2014

Sponsor: Wilson Therapeutics USA, Inc.

P.O. Box 17757 Urbana, Illinois 61803 - USA

Wilson Therapeutics, AB Västra Trädgårdsgatan 15 11453 Stockholm, Sweden

Sponsor Representative:

PD

11 Ridgefield Road Winchester, Massachusetts, 01890, USA

> Celerion 621 Rose Street Lincoln, NE 68502

### Statistical Analysis Plan Signature Page

Sponsor: Wilson Therapeutics USA, Inc. P.O. Box 17757 Urbana, Illinois 61803 - USA

> Wilson Therapeutics, AB Västra Trädgårdsgatan 15 11453 Stockholm, Sweden

Compound Name: WTX101

Protocol: WTX101-102

Study Title: A.Phase 1, Single-Center, Randomized, 3-Period Crossover Study in Healthy Volunteers to Evaluate the Absorption of WTX101 After Single Dose Administration of an Enteric Coated Formulation with and without food and a Non-Coated Formulation Coadministered with a Proton Pump Inhibitor without Food



Statistical Analysis Plan 12 May 2014


## **Table of Contents**

| 1. | | ODUCTION | |
|---|---|---|---|
| 2. | OBJE | ECTIVES AND ENDPOINTS | 4 |
| | 2.1 | Objectives | 4 |
| | 2.2 | Endpoints | |
| 3. | STU | DY DESIGN | |
| 4. | | YSIS POPULATIONS | |
| | 4.1 | Analysis Populations | 6 |
| <b>5</b> . | TREA | ATMENT DESCRIPTIONS | |
| | 5.1 | Test Treatment | |
| | 5.2 | Reference Treatment | 6 |
| 6. | PHAF | RMACOKINETIC ANALYSIS | |
| 7. | EFFI( | CACY/PHARMACODYNAMICS | 6 |
| 8. | SAFE | ETY | 7 |
| | 8.1 | Subject Discontinuation | |
| | 8.2 | Demographics | 7 |
| | 8.3 | Adverse Events | 7 |
| | 8.4 | Labs (Serum Chemistry, Hematology, Coagulation, and | |
| | | Urinalysis) | |
| | 8.5 | Vital Signs | 9 |
| | 8.6 | ECG | 9 |
| | 8.7 | Concomitant Medications | 10 |
| | 8.8 | Physical Examination | 10 |
| 9. | SUM | MARY TABLES AND FIGURES | 10 |
| 10. | | A LISTING TITLES AND NUMBERS | |
| 11. | TABL | E SHELLS | 14 |
| 12. | LISTI | NG SHELLS | 37 |

#### 1. INTRODUCTION

The following analysis plan provides the framework for the summarization of the data from this study. The analysis plan may change due to unforeseen circumstances. Any changes made after the locking of the database will be documented in the clinical study report. Please note that the header for this page will be the one used for the main body of the report.

#### 2. OBJECTIVES AND ENDPOINTS

## 2.1 Objectives

The primary objectives are:

- The effect of dosing with an Enteric coated (EC) tablet versus dosing with the current non-coated capsule administered with a proton pump inhibitor (PPI; omeprazole) under fasting conditions on the absorption of WTX101.
- The effect of dosing an EC tablet with and without food on the absorption of WTX101
- The safety and tolerability of WTX101.

## 2.2 Endpoints

The primary endpoints are:

- Plasma concentrations and PK parameters (e.g.,  $AUC_{0-inf}$ ,  $AUC_{0-inf}$ , Cmax,  $t_{max}$ ,  $\lambda_z$ , and  $t_{1/2}$ , CL/F, and Vz/F) for total Molybdenum (Mo) following WTX101 EC tablet administration under fasting and fed conditions and WTX101 non coated capsule coadministered with a PPI under fasting conditions
- Safety and tolerability will be evaluated based on physical examinations, vital sign measurements, Electrocardiogram (ECGs), adverse events (AEs), and clinical laboratory tests.

#### 3. STUDY DESIGN

This will be a single-center, open-label, randomized, 3-period, 3-treatment, 6-sequence crossover study evaluating the PK of single doses of WTX101 in healthy subjects based on the measurement of plasma total Mo.

Eighteen (18) healthy, non-tobacco using adult male and female subjects who complete the study screening assessments and meet all eligibility criteria will be enrolled. These subjects will receive the corresponding product, according to a randomization scheme generated at Celerion.

Screening of subjects will occur within 28 days prior to the first WTX101 dose.

Subjects randomized to receive PPI in Period 1 (Treatment C) will report to the Clinical Research Unit (CRU) on Day -5, i.e. 5 days prior to first dosing with WTX101, to receive a morning dose of omeprazole under fasting conditions. These subjects will be given a container with omeprazole doses and will continue once daily (QD) administration of omeprazole under fasting conditions on an outpatient basis, until their return to the CRU for check-in on Day -1. To ensure that the planned number of subjects are dosed with WTX101 on Day 1 of Period 1, stand-by subjects will also receive QD doses of omeprazole, as described above. Should any subject withdraw from the study after omeprazole administration, but before receiving WTX101 in Period 1, they will be replaced with a stand-by subject.

Subjects randomized to receive PPI in Periods 2 or 3 will receive the container with omeprazole doses prior to discharge from the CRU after the 192-hour post-dose procedures in Period 1 or Period 2, as appropriate. These subjects will initiate QD administration of omeprazole under fasting conditions at home the following day and continue until their return to the CRU for their next admission.

In each of the 3 periods, all subjects (Treatments A, B, and C) will be admitted to the CRU on Day -1, and will receive WTX101 EC tablets alone under fasting conditions (Treatment A); WTX101 EC tablets alone under fed conditions (Treatment B); or, omeprazole under fasting conditions followed by WTX101 non-coated capsules under fasting conditions (Treatment C). Pharmacokinetic (PK) sampling (for the measurement of plasma concentrations of total elemental Molybdenum (Mo)) will be obtained at the following timepoints while subjects remain in the CRU: Time 0 (within 1 hour predose), and then 1, 2, 3, 3.5, 4, 4.5, 5, 6, 7, 7.5, 8, 8.5, 9, 9.5, 10, 12, 14, 16, 24, 36, and 48 hours postdose. Subjects will be discharged on Day 3 following the 48 hours postdose procedures, unless medically necessary to extend confinement to 72 hours.

Subjects will be required to return to the CRU for outpatient visits on 6 consecutive days (Days 4, 5, 6, 7, 8 and 9) in each period, for subsequent PK sampling and procedures at: 72, 96, 120, 144, 168, and 192 hours postdose.

The washout between WTX101 doses in each period will be at least 14 days.

Subjects will return to the CRU 14 days (+/-2 days) after the final study medication administration for an end of study (EOS) visit with follow-up procedures, and to determine if any AE has occurred since the last study visit. Subjects who terminate the study early should be seen and assessed by an Investigator, whenever possible, to undergo the procedures associated with the EOS visit.

Safety will be monitored throughout the study.

Subjects who complete the study may be involved in the study for up to 48 days excluding screening (Day -5 of period one to the EOS visit).

Subjects may be replaced at the discretion of the Sponsor.

#### 4. ANALYSIS POPULATIONS

### 4.1 Analysis Populations

Safety Population: All subjects who received at least one dose of the WTX101.

### 5. TREATMENT DESCRIPTIONS

#### 5.1 Test Treatment

Treatment B: 60 mg WTX101 (2 x WTX101 EC tablets, 30mg) at Hour 0 on Day 1, 30 minutes after the start of a high-fat breakfast, preceded by an overnight fast.

Treatment C: 20 mg omeprazole (1 x 20 mg delayed-release capsule) QD on the mornings of Days -5 to -1 following an overnight fast, 20 mg omeprazole capsule at Hour -1 on Day 1 following an overnight fast, and 60 mg WTX101 (2 x WTX101 non-coated capsules, 30mg) at Hour 0 on Day 1

A brief treatment description will be used in tables and listings as:

Treatment B: 60 mg WTX101 on Day 1 (Fed).

Treatment C: 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

#### 5.2 Reference Treatment

Treatment A: 60 mg WTX101 (2 x WTX101 EC tablets, 30mg) at Hour 0 on Day 1 following an overnight fast

A brief treatment description will be used in tables and listings as:

Treatment A: 60 mg WTX101 on Day 1 (Fasted).

Treatments will be referred to in the text of the report as:

Treatment A (WTX101 alone, fasted), Treatment B (WTX101 alone, fed), and Treatment C (WTX101 with omeprazole, fasted).

### 6. PHARMACOKINETIC ANALYSIS

A separate pharmacokinetic analysis plan (PKAP) will be prepared by Kramer Consulting LLC and agreed upon with the Sponsor.

#### 7. EFFICACY/PHARMACODYNAMICS

Not applicable

#### 8. SAFETY

All clinical safety and tolerability data will be listed by subject and assessment timpoints, including rechecks, unscheduled assessments, and early termination, chronologically.

Continuous variables will be summarized using N, mean, standard deviation (SD), coefficient of variance (CV), median, minimum, and maximum. Frequency counts will be reported for all categorical data.

Decimal point will be presented as follows: N will be presented without decimal, minimum/maximum in same precision as in the database, mean/median in one more decimal than minimum/maximum, and SD in one more decimal than mean/median.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

No inferential statistics will be performed.

## 8.1 Subject Discontinuation

Individual subject's dosing status (treatment dosed) will be provided along with their completion status and date. Frequency counts of all subjects dosed in the study, completing the study, and discontinuing early from the study along with the reason for discontinuation will be tabulated by treatment sequence and overall for this presentation.

### 8.2 Demographics

Descriptive statistics will be calculated for continuous demographic variables (age, weight, height, and body mass index) and frequency counts will be tabulated for categorical demographic variables (gender, race, and ethnicity) by treatment sequence and overall.

### 8.3 Adverse Events

Adverse events (AEs) will be coded with Medical Dictionary for Regulatory Activities (MedDRA®) Version 16.1.

A treatment-emergent adverse event (TEAE) is defined as an AE that is starting or worsening at the time of or after study drug administration. An AE that occurs during the washout period between drugs is considered treatment emergent to the last drug given. If an AE that was reported during the study increases in severity that AE is given a resolution date and time and a new record initiated with the new severity. If the severity of an AE remains the same or decreases, the AE will be kept open through to resolution. All AEs captured in the database

will be listed in by-subject data listings. However, only TEAEs will be summarized. For treatment C, the TEAEs will be summarized by time interval (prior to WTX101 dosing and post WTX101 dosing) and overall.

Summary tables will include the number of subjects reporting the TEAE and percent of subjects who received study drug, number of TEAEs and percent of total TEAEs. These results will be summarized by treatment and overall. Number of subjects reporting at least one TEAE and number of TEAEs will also be summarized by treatment, severity (NCI CTCAE toxicity grading scale 5-point severity scale), and relationship to treatment. In addition, all AEs (preferred term) for all periods but exclude those who took Omeprazole in Period 1 (i.e. following first WTX101-101 dosing) will be summarized by the number and percentage of subjects with the same AE and also by severity and the relationship to drug. All AEs will be listed by subject, including verbatim term, onset date and time, resolved date and time, seriousness, severity, frequency, and relationship to treatment.

Should any serious adverse events (SAEs), AEs leading to discontinuation, and AEs resulting in death occur during this study, the AEs will be displayed in the data listings and discussed in the text of the study report.

## 8.4 Labs (Serum Chemistry, Hematology, Coagulation, and Urinalysis)

Serum chemistry, hematology, coagulation, and urinalysis will be performed at screening following a fast of at least 8 hours, the check-in for each period following a fast of at least 6 hours, 36 hour pose WTX101 dose in each period, and end of study (or upon early termination).

Descriptive statistics at specified time points (Check-in and 36 hour post WTX101 dose) will be provided for serum chemistry, hematology, coagulation, and urinalysis results by treatment. Change from Baseline [Check-in (Day -1) prior to WTX101 dosing] to the postdose time point (Hour 36) will also be provided for serum chemistry, hematology, coagulation, and urinalysis results for each treatment. Shift from baseline value tables, which provide the frequency of each shift in out of range results, will be provided by treatment for serum chemistry, hematology, coagulation, and urinalysis results. In addition, descriptive statistics at screening and end of study will be provided for serum chemistry, hematology, coagulation, and urinalysis results for all subjects as well.

All out-of-range values for serum chemistry, hematology, coagulation, and urinalysis will be listed by subject. Out-of-range values are considered to be values that are out-of normal range as defined by the clinical laboratory. The normal range values will be displayed in the data listings.

When change from baseline is calculated, baseline is the last schedule assessment before dosing of WTX101 in each period, also including rechecks and unscheduled assessments, whichever is later. Rechecks, unscheduled

assessments and early termination measurements taken after WTX101 dosing will not be used in the summarization.

Clinical laboratory values will also be displayed in a data listing by subject.

### 8.5 Vital Signs

Vital signs (blood pressure, heart rate, respiration rate, and body temperature) will be performed at screening, Check-in, predose, Hour 1, Hour 4, Hour 8, Hour 12, and Hour 24 post WTX101 dose for each period, and at the end of study (or upon early termination).

Descriptive statistics for vital sign measurements (blood pressure, heart rate, respiration rate, and body temperature) at specified time points (Check-in, predose, Hour 1, Hour 4, Hour 8, Hour 12, and Hour 24 post WTX101 dose) and change from Baseline to postdose observations will be provided for vital sign measurements by treatment. In addition, descriptive statistics at screening and end of study will be provided for vital sign measurements for all subjects as well.

When change from baseline is calculated, baseline is the last schedule assessment before dosing of WTX101 in each period, also including rechecks and unscheduled assessments, whichever is later. Rechecks, unscheduled assessments and early termination measurements taken after WTX101 dosing will not be used in the summarization.

Vital signs will also be displayed in a data listing by subject.

#### 8.6 ECG

Single 12-lead ECG will be performed at screening, Check-in, predose, Hour 1, Hour 4, Hour 8, Hour 12, and Hour 24 post WTX101 dose for each period, and at the end of study (or upon early termination).

ECGs will be performed on subjects after at least 2 minutes in supine position. All ECG tracings will be reviewed by the Study Physician or his/her designee.

Descriptive statistics will be calculated for heart rate, PR, QRS, QT, QTcB and QTcF (Bazett's and Fridericia's correction) intervals by treatment at the specified time points (Check-in, predose, Hour 1, Hour 4, Hour 8, Hour 12, and Hour 24 post WTX101 dose) as well as change from baseline to the postdose time points. In addition, descriptive statistics at screening and end of study will be provided for vital sign measurements for all subjects as well.

When change from baseline is calculated, baseline is the last schedule assessment before dosing of WTX101 in each period, also including rechecks and unscheduled assessments, whichever is later. Rechecks, unscheduled

assessments and early termination measurements taken after WTX101 dosing will not be used in the summarization.

ECG results will be classified as normal, abnormal not clinically significant, or abnormal clinically significant by the Principal Investigator (PI). Frequency of ECG results shift from baseline will be provided at specified time points by treatment.

ECGs will also be displayed in a data listing by subject.

#### 8.7 Concomitant Medications

All concomitant medications recorded during the study will be coded with the WHO Dictionary Version 01Sep2013.

## 8.8 Physical Examination

A full physical examination will be performed at screening, check-in, and at the end of the study or upon early termination. A symptom-driven physical examination may be performed at other times, at the PI's discretion. Physical examination will be presented in a data listing. A normal-abnormal shift table will also be presented for physical exam results. Abnormal findings will be discussed in the clinical study report.

#### 9. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the ICH structure. Please note that all summary tables and figures will be generated using SAS® Version 9.3 or higher.

The following is a list of table numbers and titles that will be included as summary tables:

## 14.1 Demographic Data Summary Tables

| Table 14.1.1 | Summary of Disposition |
|--------------|-------------------------|
| Table 14.1.2 | Disposition of Subjects |
| Table 14.1.3 | Demographic Summary |

## 14.2 Pharmacokinetic Data Summary Tables and Figures

Please note: This part will be covered by the separated PKAP.

## 14.3 Safety Data Summary Tables

## 14.3.1 Displays of Adverse Events

| Table 14.3.1.1 | Adverse | Event | Frequency | by | Treatment - | Number | 0 |
|---|---|---|---|---|---|---|---|
| | Subjects | Reporti | ing the Even | t (% | of Subject Dos | sed) | |

- Table 14.3.1.2 Adverse Event Frequency by Treatment Number of Adverse Events (% of Total Adverse Events)
- Table 14.3.1.3 Adverse Event Frequency by Treatment, Severity, and Relationship to Drug Number of Subjects Reporting Events
- Table 14.3.1.4 Adverse Event Frequency by Treatment, Severity, and Relationship to Drug Number of Adverse Events
- Table 14.3.1.5 Adverse Event Frequency by Severity and Relationship to Drug Following First WTX101-101 Dosing Number of Subjects Reporting Events
- Table 14.3.1.6 Adverse Event Frequency by Severity, and Relationship to Drug Following First WTX101-101 Dosing Number of Adverse Events

## 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (if no serious adverse event occurred, a statement 'No serious adverse event is reported' will be in the table.

# 14.3.3. Narratives of Deaths, other Serious and Certain other Significant Adverse Events

## 14.3.4. Abnormal Laboratory Value Listing (each patient)

- Table 14.3.4.1 Out-of-Range Values and Recheck Results Serum Chemistry
- Table 14.3.4.2 Out-of-Range Values and Recheck Results Hematology
- Table 14.3.4.3 Out-of-Range Values and Recheck Results Coagulation
- Table 14.3.4.4 Out-of-Range Values and Recheck Results Urinalysis
- Table 14.3.4.5 Out-of-Range Values and Recheck Results Other

# 14.3.5. Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

- Table 14.3.5.1 Clinical Laboratory Summary and Change from Baseline Serum Chemistry
- Table 14.3.5.2 Clinical Laboratory Shift from Baseline Serum Chemistry
- Table 14.3.5.3 Clinical Laboratory Summary and Change from Baseline Hematology
- Table 14.3.5.4 Clinical Laboratory Shift from Baseline Hematology

| Table 14.3.5.5 | Clinical Laboratory Summary and Change from Baseline – Coagulation |
|---|---|
| Table 14.3.5.6 | Clinical Laboratory Shift from Baseline – Coagulation |
| Table 14.3.5.7 | Clinical Laboratory Summary and Change from Baseline – Urinalysis |
| Table 14.3.5.8 | Clinical Laboratory Shift from Baseline – Urinalysis |
| Table 14.3.5.9 | Vital Sign Summary and Change from Baseline |
| Table 14.3.5.10 | 12-Lead Electrocardiogram Summary and Change from Baseline |
| Table 14.3.5.11 | 12-Lead Electrocardiogram Shift from Baseline |
| Table 14.3.5.12 | Physical Examination Shift from Screening |

#### 10. DATA LISTING TITLES AND NUMBERS

Note: Hepatitis and HIV results that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in any database transfer.

Data listings are numbered following the ICH structure. The following is a list of appendix numbers and titles that will be included as data listings:

## 16.1. Study Information

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

## 16.2. Subject Data Listings

## 16.2.1. Subject Discontinuation

Appendix 16.2.1 Subject Discontinuation

## 16.2.2. Protocol Deviations

Appendix 16.2.2 Protocol Deviations

## 16.2.3. Subjects Excluded from Pharmacokinetic Analysis

Appendix 16.2.3 Subjects Excluded from Pharmacokinetic Analysis

Note: Appendices 16.2.2 and 16.2.3 are generated in MS Word for inclusion in the study report

### 16.2.4. Demographic Data

Appendix 16.2.4.1 Demographics
Appendix 16.2.4.2.1 Physical Examination (I of II)
Appendix 16.2.4.2.2 Physical Examination (II of II)

| Appen | ıdix | 16 | .2.4 | 1.2.3 | Physical Examination Descriptions |
|-------|------|----|------|-------|-----------------------------------|
| _ | | | _ | | |

Appendix 16.2.4.3 Medical History
Appendix 16.2.4.4 Substance Use

## 16.2.5. Compliance and Drug Concentration Data

Appendix 16.2.5.1.1 Inclusion Criteria

Appendix 16.2.5.1.2 Exclusion Criteria

Appendix 16.2.5.2 Subject Eligibility

Appendix 16.2.5.3.1 Check-in and Return Criteria

Appendix 16.2.5.3.2 Check-in and Return Responses

Appendix 16.2.5.3.3 Check-out Date and Time

Appendix 16.2.5.4.1 Test Compound Description

Appendix 16.2.5.4.2 Test Compound Administration Times

Appendix 16.2.5.4.3 Drug and Diary Accountability

Appendix 16.2.5.5 Blood Draw Times

Appendix 16.2.5.6 Meal Times

Appendix 16.2.5.7 Concomitant Medications

### 16.2.6. Individual Pharmacokinetic Data

Please note: This part will be covered by the separated PKAP.

## 16.2.7. Individual Adverse Event Listings

Appendix 16.2.7.1 Adverse Events (I of II)

Appendix 16.2.7.2 Adverse Events (II of II)

Appendix 16.2.7.3 Adverse Event Non-Medication Procedures

Appendix 16.2.7.4 Adverse Event Preferred Term Classification

### 16.2.8. Individual Laboratory Measurements

| Appendix 16.2.8.1 | Clinical Laborator | v Report - Serum Chemistry | , |
|----------------------|----------------------|----------------------------|---|
| / NDDCHAIX TO.Z.O. I | Cili lical Eaborator | | , |

Appendix 16.2.8.2 Clinical Laboratory Report - Hematology

Appendix 16.2.8.3 Clinical Laboratory Report - Coagulation

Appendix 16.2.8.4 Clinical Laboratory Report - Urinalysis

Appendix 16.2.8.5 Clinical Laboratory Report - Urine Drug Screening

Appendix 16.2.8.6 Clinical Laboratory Report - Other

Appendix 16.2.8.7 Clinical Laboratory Report - Comments

## 16.2.9. Other Safety Observations

Appendix 16.2.9.1 Vital Signs

Appendix 16.2.9.2 12-Lead Electrocardiogram

Appendix 16.2.9.3 Phone Participant

## 11. TABLE SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables that will be included in the final report.


Table 14.1.1 Summary of Disposition

#### Treatment Sequence

| Disposition | ABC | ACB | BAC | BCA | CAB | CBA | Overall |
|---|---|---|---|---|---|---|---|
| Dosed | XX | XX | XX | XX | XX | XX | XX |
| Completed | XX | XX | XX | XX | XX | XX | XX |
| Discontinued Early | X | X | X | X | X | X | X |
| <discontinuation reason=""></discontinuation> | X | X | X | X | X | X | X |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM


Table 14.1.2 Disposition of Subjects

| Randomized | | Treatment Dosed | | | | | pleted | Study Completion | |
|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Dosing<br>Sequence | A | В | C A B C | | Status | Date | | |
| X | XXX | Yes | Yes | Yes | Yes | Yes | Yes | Completed Study | DDMMYYYY |
| X | XXX | No | Yes | Yes | No | Yes | Yes | Terminated Study Prematurely | DDMMYYYY |
| X | XXX | Yes | Yes | Yes | Yes | Yes | Yes | Completed Study | DDMMYYYY |
| X | XXX | Yes | Yes | Yes | Yes | Yes | Yes | Completed Study | DDMMYYYYY |
| X | XXX | Yes | Yes | Yes | Yes | Yes | Yes | Completed Study | DDMMYYYY |
| X | XXX | Yes | Yes | Yes | Yes | Yes | Yes | Completed Study | DDMMYYYY |
| XX | XXX | Yes | Yes | Yes | Yes | Yes | Yes | Terminated Study Prematurely | DDMMYYYY |
| XX | XXX | Yes | Yes | Yes | Yes | Yes | Yes | Completed Study | DDMMYYYY |
| | | XX | XX | XX | XX | XX | XX | | |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYY HH:MM


Table 14.1.3 Demographic Summary

#### Treatment Sequence

| Trait | | ABC | ACB | BAC | BCA | CAB | CBA | Overall |
|---|---|---|---|---|---|---|---|---|
| <br>Gender | Female | XX | XX | XX | XX | XX | XX | XX |
| | Male | XX | XX | XX | XX | XX | XX | XX |
| Race | White | XX | XX | XX | XX | XX | XX | XX |
| | Black or African American | XX | XX | XX | XX | XX | XX | XX |
| | Asia | XX | XX | XX | XX | XX | XX | XX |
| Ethnicity | Hispanic or Latino | XX | XX | XX | XX | XX | XX | XX |
| _ | Not Hispanic or Latino | XX | XX | XX | XX | XX | XX | XX |
| Age | N | Х | X | X | X | Х | X | X |
| - | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | CV | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM


Table 14.1.3 Demographic Summary

#### Treatment Sequence

| Trait | | ABC | ACB | BAC | BCA | CAB | CBA | Overall |
|---|---|---|---|---|---|---|---|---|
| Weight (kg) | N | Х | X | X | X | X | X | X |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | CV | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Height (cm) | N | X | X | X | X | Х | X | X |
| - | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | CV | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Body Mass Index (kg | g/m²) N | X | X | X | X | X | Х | X |
| - | Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | CV | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYY HH:MM


Table 14.3.1.1 Adverse Event Frequency by Treatment - Number of Subjects Reporting Events (% of Subjects Dosed)

| | | | Treat | ment | | | |
|---|---|---|---|---|---|---|---|
| | | | | С | | Overall Following | |
| Adverse Event* | A | В | Prior to<br>WTX101<br>Dosing | Post<br>WTX101<br>Dosing | Overall | the First WTX101 Dosing | Overall |
| Number of Subjects Dosed<br>Number of Subjects With Adverse Events<br>Number of Subjects Without Adverse Events | XX (100%)<br>X ( XX%)<br>X ( XX%) | XX (100%)<br>X ( XX%)<br>X ( XX%) | XX (100%)<br>X ( XX%)<br>X ( XX%) | XX (100%)<br>X ( XX%)<br>X ( XX%) | XX (100%)<br>X ( XX%)<br>X ( XX%) | XX (100%)<br>X ( XX%)<br>X ( XX%) | XX (100%)<br>X ( XX%)<br>X ( XX%) |
| System Organ Class Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term Preferred Term | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%) | X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) |

Note: \* Adverse events are classified according to MedDRA Version 16.1. Each Subject was only counted once per preferred term.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM


Table 14.3.1.2 Adverse Event Frequency by Treatment - Number of Adverse Events (% of Total Adverse Events)

| | | | C | | | Overall | |
|---|---|---|---|---|---|---|---|
| Adverse Event* | A | В | Prior to Post<br>WTX101 WTX101<br>Dosing Dosing | | Overall | Following<br>the First<br>WTX101<br>Dosing | Overall |
| Number of Adverse Events | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| System Organ Class | | | | | | | |
| Preferred Term | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Preferred Term | X ( X%) | x ( x%) | x ( x%) | x ( x%) | x ( x%) | x ( x%) | X ( X%) |

Note: \* Adverse events are classified according to MedDRA Version 16.1.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas prg/stsas/tab PROGRAMNAME.sas DDMMYYYY HH:MM

Table 14.3.1.3 Adverse Event Frequency by Treatment, Severity, and Relationship to Drug
- Number of Subjects Reporting Events

| | Number of<br>Subjects with | Severity Grade | | | | | Relationship to Drug | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Treatment | Adverse Events | 1 | 2 | 3 | 4 | 5 | Likely | Probably | Possibly | Unlikely | Unrelated |
| Abdominal pain | А | X | Χ | Х | Х | Х | Х | X | X | X | X | X |
| Constipation | A | X | X | X | X | X | X | X | X | X | X | X |
| Headache | A | X | X | X | X | X | X | X | X | X | X | X |
| | В | X | X | X | X | X | X | X | X | X | X | X |
| Myalgia | A | X | X | X | X | X | X | X | X | X | X | X |
| Nasal congestion | n C1 | X | X | X | X | X | X | X | X | X | X | X |
| Skin laceration | C2 | X | X | X | Х | X | Х | X | X | X | X | X |
| Treatment A | | X | Х | X | Х | Х | Х | Х | X | X | X | X |
| Treatment B | | X | X | X | X | X | X | X | X | X | X | X |
| Treatment C1 | | X | X | X | X | X | X | X | X | X | X | X |
| Treatment C2 | | X | X | X | X | X | X | X | X | X | X | X |
| Treatment C | | X | Χ | Χ | X | Χ | X | X | X | X | X | X |
| Overall | | X | Х | Х | X<br> | X<br> | Х | X | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 16.1.

When a subject experienced the same AE at more than one level of severity during a treatment period, only the most severe one was counted. When a subject experienced the same AE at more than one level of drug relationship during a treatment period, only the most related one was counted.

Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Death due to AE.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Treatment C1 = Treatment C prior to WTX101 dosing, Treatment C2 = Treatment C post WTX101 dosing

Program: /AAXXXXX/ECR/sas prg/stsas/tab tblae3a auto.sas DDMMMYYYY HH:MM


Table 14.3.1.4 Adverse Event Frequency by Treatment, Severity, and Relationship to Drug
- Number of Adverse Events

| | | Number of | | Seve | erity | Grade | : | | Rela | tionship | to Drug | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Treatment | Adverse Events | 1 | 2 | 3 | 4 | 5 | Likely | Probably | Possibly | Unlikely | Unrelated |
| Abdominal pain | А | X | Х | Х | Х | Х | Х | X | Х | X | Х | X |
| Constipation | A | X | X | X | X | X | X | X | X | X | X | X |
| Headache | A | X | X | X | X | X | X | X | X | X | X | X |
| | В | X | X | X | X | X | X | X | X | X | X | X |
| Myalgia | A | X | X | Χ | X | X | X | X | X | X | X | X |
| Nasal congestion | C1 | X | X | Χ | X | X | X | X | X | X | X | X |
| Skin laceration | C2 | Х | Х | Х | X | X | Х | X | X | X | X | X |
| Treatment A | | X | Х | Х | Х | X | Х | X | X | X | X | X |
| Treatment B | | X | Χ | X | X | X | X | X | X | X | X | X |
| Treatment C1 | | X | X | Χ | X | X | X | X | X | X | X | X |
| Treatment C2 | | X | Χ | X | X | X | X | X | X | X | X | X |
| Treatment C | | X | Χ | X | X | X | X | X | X | X | X | X |
| Overall | | X | Χ | Χ | Χ | Χ | Χ | X | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 16.1.

Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Death due to AE.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Treatment C1 = Treatment C prior to WTX101 dosing, Treatment C2 = Treatment C post WTX101 dosing

Program: /AAXXXXX/ECR/sas prg/stsas/tab tblae4a auto.sas DDMMMYYYY HH:MM


Table 14.3.1.5 Adverse Event Frequency by Severity and Relationship to Drug Following First WTX101-101 Dosing
- Number of Subjects Reporting Events

| | Number of<br>Subjects with | Severity Grade | | | | | Relationship to Drug | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Adverse Events | 1 | 2 | 3 | 4 | 5 | Likely | Probably | Possibly | Unlikely | Unrelated |
| Abdominal pain | Х | X | X | Х | Х | X | X | X | X | X | X |
| Constipation | X | X | X | X | X | X | X | X | X | X | X |
| Headache | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X |
| Myalgia | X | X | X | X | X | X | X | X | X | X | X |
| Nasal congestion | X | X | X | X | X | X | X | X | X | X | X |
| Skin laceration | X | Χ | Χ | Χ | Χ | Χ | X | X | X | X | X |
| Overall | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

Note: \* Adverse events are classified according to MedDRA Version 16.1.

When a subject experienced the same AE at more than one level of severity during a treatment period, only the most severe one was counted. When a subject experienced the same AE at more than one level of drug relationship during a treatment period, only the most related one was counted.

Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Death due to AE.

Program: /AAXXXXX/ECR/sas prg/stsas/tab tblae3a auto.sas DDMMMYYYY HH:MM


Table 14.3.1.6 Adverse Event Frequency by Severity and Relationship to Drug Following First WTX101-101 Dosing
- Number of Adverse Events

| | Number of | Severity Grade | | | | | Relationship to Drug | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Event* | Adverse Events | 1 | 2 | 3 | 4 | 5 | Likely | Probably | Possibly | Unlikely | Unrelated |
| Abdominal pain | X | Х | X | X | Х | Х | X | Х | Х | X | Х |
| Constipation | X | X | X | X | X | X | X | X | X | X | X |
| Headache | X | X | X | X | X | X | X | X | X | X | X |
| | X | X | X | X | X | X | X | X | X | X | X |
| Myalgia | X | X | X | X | X | X | X | X | X | X | X |
| Nasal congestion | X | X | X | X | X | X | X | X | X | X | X |
| Skin laceration | Х | X | X | X | X | X | X | X | X | Х | X |
| Overall | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х |

Note: \* Adverse events are classified according to MedDRA Version 16.1.

Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Death due to AE.

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab tblae4a\_auto.sas DDMMMYYYY HH:MM

Wilson Therapeutics USA, Inc. WTX101: WTX101-102 Celerion, Clinical Study Report No. CA13895


Table 14.3.2.1 Serious Adverse Events

\_\_\_\_\_

No serious adverse event is reported during the study.

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab cdash\_tblae\_ser.sas DDMMYYYY HH:MM


Table 14.3.4.1 Out-of-Range Values and Recheck Results - Serum Chemistry

| Subject Age/<br>Number Gender | Study<br>Period | Treatment | Day | Hour | Date | Test Name<br>X.X-XX.X<br>(mg/dL) | Test Name<br>X.X-X.X<br>(mEq/L) | Test Name<br>XXX-XXX<br>(mEq/L) | Test Name<br>X.X-X<br>(g/dL) | Test Name<br>F: X-XX<br>M: X-XX<br>(mg/dL) |
|---|---|---|---|---|---|---|---|---|---|---|
| X XX/M | Screen | | | | DDMMYYYY | X.X | X.X LN | XXX | X.X | XX |
| | 1 | A | -X | -X.X | DDMMYYYY | X.X | X.X LN | XXX | X.X | XX |
| | | | X | X.X | DDMMYYYY | X.X | X.X LN | XXX | X.X | XX |
| | 2 | В | -X | -X.X | DDMMYYYY | X.X | X.X LN | XXX | X.X | XX |
| | | | X | X.X | DDMMYYYYY | X.X | X.X LN | XXX | X.X | XX |

Note: H = Above Normal Range, L = Below Normal Range

Computer: N = Not Clinically Significant, Y = Clinically Significant

PI interpretation: - = Not Clinically Significant Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Please note that Table 14.3.4.2-5 will resemble 14.3.4.1.

Page 1 of X Table 14.3.5.1 Clinical Laboratory Summary and Change From Baseline - Serum Chemistry

| | Treatment | | | Change 1 | From Basel: | ine | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test (unit) | Normal Range | Time point | Statistic | Overall | A | В | С | A | В | C |
| Test Name (unit) | XX.X - XX.X | Screen | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | | | | | | |
| | | Baseline | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | | | |
| | | Hour 36 | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XXX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX |
| | | End of Study | N Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | | | | | | |

<Similar for remaining tests.>

Note: Baseline is the last observation, including rechecks, obtained prior to dosing of WTX101 in the treatment period.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYYY HH:MM

Please note that Tables 14.3.5.3, 14.3.5.5, and 14.3.5.7 will resemble 14.3.5.1.

Celerion, Clinical Study Report No. CA13895


Table 14.3.5.2 Clinical Laboratory Shift From Baseline - Serum Chemistry

| | | | | | Baseline* 1 | L | | Baseline* N | 1 | 1 | Baseline* H | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Marmal | | | | Postdose | | | Postdose | | | Postdose | |
| Laboratory Test | Normal<br>Range | Time Point | Treat-<br>ment | L | N | Н | | N | Н | | N | Н |
| Test Name (units) | XX-XXX | Hour 36 | A<br>B<br>C | X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%)<br>XX ( XX%)<br>XX ( XX%) | X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%)<br>XX ( XX%)<br>XX ( XX%) | X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%)<br>XX ( XX%)<br>XX ( XX%) | X ( X%)<br>X ( X%)<br>X ( X%) |

<Similar for remaining laboratory tests and time points>

Note: L = Below Normal Range, N = Within Normal Range, H = Above Normal Range.

\* Baseline is the last observation, including rechecks, obtained prior to dosing of WTX101 in the treatment period.

The percentage are based on the number of subjects within the test\*treatment\*timepoint.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas prg/stsas/tab PROGRAMNAME.sas DDMMMYYYY HH:MM

Please note that Tables 14.3.5.4 and 14.3.5.6 will resemble 14.3.5.2.


Table 14.3.5.8 Clinical Laboratory Shift From Baseline - Urinalysis

| | | | | ine* N | Baseline* O | | |
|---|---|---|---|---|---|---|---|
| | 27 | | | Post | .dose | Post | dose |
| Laboratory Test | Normal<br>Range | Time Point | Treatment | N | 0 | N | 0 |
| Test Name (units) | XX-XXX | Hour 36 | А<br>В<br>С | X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%) |

<Similar for remaining laboratory tests and time points>

Note: N = Within Normal Range, O = Outside Normal Range.

\* Baseline is the last observation, including rechecks, obtained prior to dosing of WTX101 in the treatment period.

The percentage are based on the number of subjects within the test\*treatment\*timepoint.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Table 14.3.5.9 Vital Sign Summary and Change From Baseline

| | | | | Т | reatment | | Change F | rom Baseli | ne |
|---|---|---|---|---|---|---|---|---|---|
| Measurement (unit) | Time point | Statistic | Overall | A | В | C | A | В | C |
| Test Name (unit) | Screen | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | | | | | | |
| | Check-in | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XXX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | | | |
| | Baseline | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XXX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | | | |
| | Hour 1 | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | | XX<br>X.XX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.X |

<Similar for remaining time points and measurements. For the end of study time point, all subjects will be pooled together as overall as for screen time point.>

Note: Baseline is the last observation, including rechecks, obtained prior to dosing of WTX101 in the treatment period. Treatment A = 60 mg WTX101 on Day 1 (Fasted)


WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)


Table 14.3.5.10 12-Lead Electrocardiogram Summary and Change From Baseline

| | | | | T | reatment | | Change F | rom Baseli | ne |
|---|---|---|---|---|---|---|---|---|---|
| Parameter (unit) | Time point | Statistic | Overall | A | В | С | A | В | C |
| Heart Rate (bpm) | Screen | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | | | | | | |
| | Check-in | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | | | |
| | Baseline | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | | | |
| | Hour 1 | N<br>Mean<br>SD<br>CV<br>Median<br>Minimum<br>Maximum | | XX<br>X.XX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX<br>X.X | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX | XX<br>X.XX<br>X.XXX<br>X.XXX<br>X.XX<br>X.XX |

<Similar for remaining time points and parameters. For the end of study time point, all subjects will be pooled together as overall as for screen time point.>

Note: Baseline is the last non-missing measurement, including rechecks, obtained prior to dosing of WTX101 in the treatment period. Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)


Table 14.3.5.11 12-Lead Electrocardiogram Shift From Baseline

| | | Baseline = N Baseline = ANCS | | NCS | Ва | seline = A | ACS | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Postdose | | Postdose | | | Postdos | se |
| Treatment | Time Point | N | ANCS A | CS N | ANCS | ACS | N | ANCS | ACS |
| A | Hour 1<br>Hour 4<br>Hour 8<br>Hour 12<br>Hour 24 | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%) X ( XX ( XX%) X ( XX ( XX%) X ( XX%) X ( XX%) X ( XX%) X ( XX ( X | X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( | X%) XX ( XX%)<br>X%) XX ( XX%)<br>X%) XX ( XX%) | X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%)<br>XX ( XX%)<br>XX ( XX%)<br>XX ( XX%)<br>XX ( XX%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) |
| В | Hour 1<br>Hour 4<br>Hour 8<br>Hour 12<br>Hour 24 | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%) X ( XX ( XX%) X ( XX ( XX%) X ( XX%) X ( XX ( X | X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( | X%) XX ( XX%)<br>X%) XX ( XX%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%)<br>XX ( XX%)<br>XX ( XX%)<br>XX ( XX%)<br>XX ( XX%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) |
| С | Hour 1<br>Hour 4<br>Hour 8<br>Hour 12<br>Hour 24 | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%) X ( XX ( XX%) X ( XX ( XX%) X ( XX%) X ( XX%) X ( XX ( X | X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( X%) X ( | X%) XX ( XX%)<br>X%) XX ( XX%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) | XX ( XX%)<br>XX ( XX%)<br>XX ( XX%)<br>XX ( XX%)<br>XX ( XX%) | X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%)<br>X ( X%) |

Note: N = Normal, ANCS = Abnormal, Not Clinically Significant, ACS = Abnormal, Clinically Significant

Baseline is last non-missing measurements, including rechecks, obtained prior to dosing of WTX101 in the treatment period.

Percentages are based on total number of observations for each treatment at each time point.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole  $Q\bar{D}$  on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Program: /AAXXXXX/ECR/sas prg/stsas/tab ecgshift.sas DDMMMYYYY HH:MM


Table 14.3.5.12 Physical Examination Shift From Screening

| | | Screen = Normal | | Screen = A | bnormal |
|---|---|---|---|---|---|
| | | Durin | ng Study | During | Study |
| System | Time Point | Normal | Abnormal | Normal | Abnormal |
| XXXXXXX | Period 1 Check-in | Х | X | X | X |
| | Period 2 Check-in | X | X | X | X |
| | Period 3 Check-in | X | X | X | X |
| | End of Study | X | X | X | X |
| XXXXXXX | Period 1 Check-in | X | X | X | X |
| | Period 2 Check-in | X | X | X | X |
| | Period 3 Check-in | X | X | X | X |
| | End of Study | X | X | X | X |
| XXXXXXX | Period 1 Check-in | X | X | X | X |
| | Period 2 Check-in | X | X | X | X |
| | Period 3 Check-in | X | X | X | X |
| | End of Study | X | X | X | X |

Program: /AAXXXXX/ECR/sas\_prg/stsas/tab ecgshift.sas DDMMMYYYY HH:MM

Wilson Therapeutics USA, Inc. WTX101: WTX101-102 Celerion, Clinical Study Report No. CA13895

## **12. LISTING SHELLS**

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be included in the final report.


Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

| Laboratory Group | Test Name | Gender | Age Category | Normal Range | Unit |
|---|---|---|---|---|---|
| Serum Chemistry | Test Name | | $\Leftrightarrow$ | XX - XX | units |
| _ | Test Name | <> | $\Leftrightarrow$ | XX - XX | units |
| | Test Name | $\Leftrightarrow$ | $\Leftrightarrow$ | XX - XX | units |
| | Test Name | <> | $\Leftrightarrow$ | XX - XX | units |
| | Test Name | <> | $\Leftrightarrow$ | XX - XX | units |
| | Test Name | $\Diamond$ | $\Leftrightarrow$ | XX - XX | units |
| Hematology | Test Name | $\Diamond$ | $\Leftrightarrow$ | xx - xx | units |
| | Test Name | <> | $\Leftrightarrow$ | XX - XX | units |

<similar for remaining Laboratory Groups and Test Names>


Appendix 16.2.1 Subject Discontinuation

| | Subject<br>Number | Study<br>Period | Date | Completed<br>Study? | Reason for Discontinuation Comment |
|---|---|---|---|---|---|
| _ | Х | Post | DDMMYYYYY | Yes | |
| | X | Post | DDMMYYYYY | Yes | |
| | X | Post | DDMMYYYYY | Yes | |
| | X | Post | DDMMYYYY | Yes | |
| | X | Post | DDMMYYYY | No | Personal Reason |
| | X | Post | DDMMYYYYY | Yes | |
| | X | Post | DDMMYYYYY | Yes | |
| | X | Post | DDMMYYYYY | Yes | |

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895

### Appendix 16.2.4.1 Demographics


| Subject<br>Number | Date Of<br>Birth | Age<br>(yrs) | Gender | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m^2) | Informed<br>Consent<br>Date |
|---|---|---|---|---|---|---|---|---|---|
| X | DDMMYYYY | XX | XXXX | XXXXXXXXX | XXXXXXXXXX | XX.X | XXX.X | XX.XX | DDMMYYYY |
| X | DDMMYYYYY | XX | XXXX | XXXXXXXX | XXXXXXXXXX | XX.X | XXX.X | XX.XX | DDMMYYYYY |
| X | DDMMYYYY | XX | XXXX | XXXXXXXXX | XXXXXXXXXX | XX.X | XXX.X | XX.XX | DDMMYYYYY |
| X | DDMMYYYYY | XX | XXXX | XXXXXXXXX | XXXXXXXXXXX | XX.X | XXX.X | XX.XX | DDMMYYYYY |

## Celerion, Clinical Study Report No. CA13895


#### Appendix 16.2.4.2.1 Physical Examination (I of II)

| Subject<br>Number | Study<br>Period | Day | Hour | Date | Was PE<br>Performed? | System1 | System2 | System3 | System4 | System5 |
|---|---|---|---|---|---|---|---|---|---|---|
| X | Screen<br>X | X | X | DDMMYYYY<br>DDMMYYYYY | 120 | NORMAL<br>NORMAL | NORMAL<br>NORMAL | NORMAL<br>NORMAL | NORMAL<br>NORMAL | NORMAL<br>NORMAL |

Note: \* = See Appendix 16.2.4.2.3 Physical Examination Description. HEENT = Head, Eyes, Ears, Nose, Throat.

## Celerion, Clinical Study Report No. CA13895


Appendix 16.2.4.2.2 Physical Examination (II of II)

| Subject<br>Number | Study<br>Period | Day | Hour | Date | System6 | System7 | System8 | System9 | Etc. |
|---|---|---|---|---|---|---|---|---|---|
| X | Screen<br>x | · × | • | DDMMYYYY<br>DDMMWYYYY | NORMAL<br>NORMAL | NORMAL<br>NORMAL | NORMAL<br>NORMAL | NORMAL<br>NORMAL | NORMAL<br>NORMAI |

Note: \* = See Appendix 16.2.4.2.3 Physical Examination Descriptions.

Celerion, Clinical Study Report No. CA13895

### Appendix 16.2.4.2.3 Physical Examination Descriptions

|------|----|-----|
| raye | OT | - 4 |

| Subject<br>Number | Study<br>Period | Day | Hour | Date | Result | System | Description or Comment |
|---|---|---|---|---|---|---|---|
| X | Screen | • | • | DDMMYYYY | ABNORMAL | Skin | RIGHT CHEST SCAR-NCS |
| X | Screen | | • | DDMMYYYY | ABNORMAL | Skin | ABDOMINAL SCAR-NCS |
| X | Screen | • | | DDMMYYYY | ABNORMAL | Skin | ABDOMINAL SCAR-NCS |
| XX | Χ | Х | X | DDMMYYYY | ABNORMAL | Skin | ABDOMINAL SCAR-NCS |
| XX | Screen | | | DDMMYYYY | ABNORMAL | Back | MILD SCOLIOSIS-NCS |

Note: HEENT = Head, Eyes, Ears, Nose, Throat, NCS = Not Clinically Significant.

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895


### Appendix 16.2.4.3 Medical History

| | | | | | Date | | | |
|---|---|---|---|---|---|---|---|---|
| _ | | Study<br>Period | System Reviewed | Category | Start | End | Ongoing? | Condition or Event |
| X | XXX | Screen | XXXXXX XXXXX | Medical<br>Surgical | DDMMYYYY<br>DDMMYYYY | DDMMYYYY | YES<br>NO | XXXXXXX XXXXXXX XXXXXXXX |
| X | XXX | Screen | XXXXXXX XXXXX | Medical | DDMMYYYY | DDMMYYYY | NO | |

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895


### Appendix 16.2.4.4 Substance Use

| Subject<br>Number | | Substance | Description of Use | Start<br>Date | End<br>Date | Description |
|---|---|---|---|---|---|---|
| X | Screen | xxxxxxx xxx | XXXXX XXXXXXX XXXXXX | MMYYYY | <added date="" different="" end="" from="" if="" is="" start=""></added> | XXXXXXXXX XXXXX XXXX |

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895


Appendix 16.2.5.1.1 Inclusion Criteria

X. <>?

Appendix 16.2.5.1.2 Exclusion Criteria


WTX101: WTX101-102

## Celerion, Clinical Study Report No. CA13895


### Appendix 16.2.5.2 Subject Eligibility

| Subject<br>Number | Study<br>Period | Did subject meet all eligibility criteria? | Criterion Not Met* | Specify |
|---|---|---|---|---|
| X | Screen | No | EXCLUSION X | XXXXXXXXXXXXXX XXXX |
| X | Screen | Yes | | |
| X | Screen | Yes | | |
| X | Screen | No | INCLUSION X | XXXXXXXXX XXXXXXXX |

Note: \* = Please refer to Appendices 16.2.5.1.1 and 16.2.5.1.2 for specific inclusion and exclusion criteria.


Appendix 16.2.5.3.1 Check-in and Return Criteria

X. < >?

X. IF (Y)ES TO ANY QUESTION, WAS SUBJECT APPROVED FOR STUDY?

## Celerion, Clinical Study Report No. CA13895


Appendix 16.2.5.3.2 Check-in and Return Responses

| | ~. 1 | | Check-in Criteria | |
|---|---|---|---|---|
| Subject<br>Number | Study<br>Period | Date | X X | Comment |
| X | X<br>X<br>X | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | No N/A<br>No N/A<br>No N/A | Will only be present and populated if there is a comment present in the study database. |
| X | X<br>X<br>X | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | No N/A<br>No N/A<br>No N/A | |
| X | X<br>X<br>X | DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY | No N/A<br>No N/A<br>No N/A | |

Note: N/A = Not Applicable.

WTX101: WTX101-102

# Celerion, Clinical Study Report No. CA13895


Appendix 16.2.5.3.3 Check-out Date and Time

| ~ 1 ! . | ~. · | Check-out | | |
|-------------------|-----------------|-----------|-------|---------|
| Subject<br>Number | Study<br>Period | Date | Time | Comment |
| X | X | DDMMYYYY | HH:MM | |
| | X | DDMMYYYY | HH:MM | |
| | X | DDMMYYYY | HH:MM | |
| X | X | DDMMYYYY | HH:MM | |
| | X | DDMMYYYY | HH:MM | |
| | X | DDMMYYYY | HH:MM | |
| X | X | DDMMYYYY | HH:MM | |
| | X | DDMMYYYY | HH:MM | |
| | X | DDMMYYYYY | HH:MM | |

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895

Appendix 16.2.5.4.1 Test Compound Description

| Compound | Form | Route |
|-------------|------|-------|
| XXXXXXXXXXX | < > | XXXX |
| YYYYYYYYYY | < > | XXXX |

Program: /AAXXXXX/ECR/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM


Celerion, Clinical Study Report No. CA13895

Appendix 16.2.5.4.2 Test Compound Administration Times

| Page | 1 | of | V |
|------|---|----|---|
| rage | | OT | Λ |

| Subject<br>Number | Study<br>Period | Treatment | Day | Hour | Date | Actual<br>Time | Compound | Dos | sage | Did You<br>Fast? | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Χ | X | X | X | х.х | DDMMYYYY | X:XX:XX | XXXXXXXXX | < > | > | XXX | |
| | X | X | X | X.X | DD <b>MM</b> MYYYY | X:XX:XX | XXXXXXXX | < > | > | XXX | |
| | X | X | X | X.X | DDMMYYYYY | X:XX:XX | XXXXXXXX | < > | > | XXX | |
| | | X | X | X.X | DDMMYYYYY | X:XX:XX | XXXXXXXX | < > | > | XXX | |
| | | X | X | X X | DDMMMYYYY | X • XX • XX | XXXXXXXXX | < > | > | XXX | |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

WTX101: WTX101-102

### Celerion, Clinical Study Report No. CA13895

Appendix 16.2.5.4.3 Drug and Diary Accountability

| Subject<br>Number | Study<br>Period | Date | Time | (1)<br>Diary? | If no, (2) Dispense Test<br>Comment Compounds? | (3) Condition of Test Compound<br>Turn in Diary? | /<br>Treatment | Comments |
|---|---|---|---|---|---|---|---|---|
| X | ALL | DDMMYYYY | X:XX:XX | XXX | XXX | XXX | X | |
| X | ALL | DDMMYYYY | X:XX:XX | XXX | XXX | XXX | X | |
| X | AT.T. | DDMMMYYYY | x • x x • x x | XXX | XXX | XXX | × | |

Note: (1) Was the subject given the test compound, dosing diary and instructions?

Program: /AAXXXXX/ECR/sas prg/stsas/lis PROGRAMNAME.sas DDMMYYYY HH:MM


<sup>(2)</sup> Was the subject instructed to take the doses as directed on the drug packaging at their scheduled time with 240 mL of water?

<sup>(3)</sup> Did the subject return their diary and test compound container (empty or not)?

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

## Celerion, Clinical Study Report No. CA13895


#### Appendix 16.2.5.5 Blood Draw Times

| Subject<br>Number | Study<br>Period | Treatment | Day | Hour | Date | Actual<br>Time | Bioassay Comments |
|---|---|---|---|---|---|---|---|
| X | X | X | Х | -X.XX | DDMMYYYY | X:XX:XX | XXXXXXXXX |
| | | | | X.XX | DDMMYYYYY | X:XX:XX | XXXXXXXXX |
| | | | | X.XX | DDMMYYYY | X:XX:XX | XXXXXXXXX |
| | | | | X.XX | DDMMYYYYY | XX:XX:XX | XXXXXXXXX |
| | | | | X.XX | DDMMYYYYY | XX:XX:XX | XXXXXXXXX |
| | | | | X.XX | DDMMYYYY | XX:XX:XX | XXXXXXXXX |
| | | | | X.XX | DDMMYYYY | XX:XX:XX | XXXXXXXXX |
| | | | | XX.XX | DDMMYYYY | XX:XX:XX | XXXXXXXXX |
| | | | | XX.XX | DDMMYYYY | XX:XX:XX | XXXXXXXXX |
| | | | X | XX.XX | DDMMYYYY | X:XX:XX | XXXXXXXXX |
| | | | | XX.XX | DDMMYYYY | X:XX:XX | XXXXXXXXX |
| | | | | XX.XX | DDMMYYYY | XX:XX:XX | XXXXXXXXX |
| | | | X | XX.XX | DDMMYYYYY | X:XX:XX | XXXXXXXXX |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Celerion, Clinical Study Report No. CA13895

### Appendix 16.2.5.6 Meal Times


| Subject<br>Number | | Treatment | Day | Hour | Event | Date | Start<br>Time | Stop<br>Time | Time Interval<br>(Start HR to Stop HR) | Comments |
|---|---|---|---|---|---|---|---|---|---|---|
| Х | X | X | -X<br>X | X.X | | DDMMYYYY | XX:XX:XX | XX:XX:XX | X.X to X.X | |
| | | | | X.X | LUNCH<br>DINNER<br>SNACK | DDMMYYYY<br>DDMMYYYY<br>DDMMYYYY | XX:XX:XX<br>XX:XX:XX<br>XX:XX:XX | XX:XX:XX | | |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

WTX101: WTX101-102

## Celerion, Clinical Study Report No. CA13895

Appendix 16.2.5.7 Concomitant Medications


| Subject<br>Number | | | Medication<br>(WHO* Term) | Dosage | Route | Start<br>Date | Start<br>Time | Stop<br>Date | Stop<br>Time E | requency | Indication | Continuing? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| X | Screen<br>1 | X | None<br>ACETAMINOPHEN<br>(ACETAMINOPHEN) | 620 mg | ORAL | DDMMYYYY | Y HH:MM | HH:MM | DDMMYYY | MY Once | Toothache | No |

Note: Concomitant medications are coded with WHO Dictionary Version 01SEP2013.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

## Celerion, Clinical Study Report No. CA13895


#### Appendix 16.2.7.1 Adverse Events (I of II)

| 2.1. | QL 1 | | | | | Time from Last Dose Onset | | | Resolved | Ė | Duration |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Period: | | | Adverse Event* | Preferred Term | (DD:HH:MM) | Date | Time | Date | Time | (DD:HH:MM) |
| PPD | Screen<br>1 | Х | Yes | None<br>XXXXXXXXXXXX | ************************************** | xx:xx:xx | DDMMYYYY | X:XX I | DDMMYYYY | x:xx | xx:xx:xx |

Note: ^ = Abbreviation for treatment-emergent, \* = Adverse events are classified according to the MedDRA Version 16.1.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Treatment C1 = Treatment C prior to WTX101 dosing, Treatment C2 = Treatment C post WTX101 dosing

Program: /AAXXXXX/ECR/sas prg/stsas/lis PROGRAMNAME.sas DDMMMYYYY HH:MM

### Celerion, Clinical Study Report No. CA13895

Appendix 16.2.7.2 Adverse Events (II of II)


| Subject | Study | | Adverse | Onset | ;<br> | | | | | Relation-<br>ship to<br>Study | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Treatment | | Date | Time | Freq | Severit | y Ser* | Outcome | Drug | Action |
| PPD | Screen<br>1 | X | None<br>XXXXXXXXXXXXXXXXXXXXXXXX | DDMMYYYY | x:xx | Inter. | <br>Grade 1 | <br>NS | Resolved | | None |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Treatment C1 = Treatment C prior to WTX101 dosing, Treatment C2 = Treatment C post WTX101 dosing

Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Death due to AE.

Ser\* represents Serious: NS = Not Serious

Freq represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous

Program: /AAXXXXX/ECR/sas prg/stsas/lis PROGRAMNAME.sas DDMMMYYYY HH:MM

## Celerion, Clinical Study Report No. CA13895


Appendix 16.2.7.3 Adverse Event Non-Medication Procedures

| Subject Study | | | Adverse | Onset<br> | | Pro | cedure | Given |
|---|---|---|---|---|---|---|---|---|
| | | Treatment | | Date | Time | Date | Time | Description |
| Х | Х | X | DRY LIPS | DDMMYYYY | XX:XX | DDMMYYYY | XX:XX | PETROLEUM JELLY |
| X | X | X | CONSTIPATION | DDMMYYYY | XX:XX | DDMMYYYY | XX:XX | PRUNE JUICE |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Treatment C1 = Treatment C prior to WTX101 dosing, Treatment C2 = Treatment C post WTX101 dosing

Program: /AAXXXXX/ECR/sas prg/stsas/lis PROGRAMNAME.sas DDMMMYYYY HH:MM

### WTX101: WTX101-102

## Celerion, Clinical Study Report No. CA13895


#### Appendix 16.2.7.4 Adverse Event Preferred Term Classification

| | | | | | | Unset | _ |
|---|---|---|---|---|---|---|---|
| Subject | Study | Adverse | | | | | |
| Number | , = | | | Preferred Term | Body System | Date | Time |
| PPD | 1 X | XXXXXXX | XXXXX XXXX XXXXX | XXXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXX | DDMMYYYY<br>DDMMYYYYY | X:XX |

Note: \* Adverse events are classified according to the MedDRA Version 16.1.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

Treatment C1 = Treatment C prior to WTX101 dosing, Treatment C2 = Treatment C post WTX101 dosing

Program: /AAXXXXX/ECR/sas prg/stsas/lis PROGRAMNAME.sas DDMMMYYYY HH:MM

Celerion, Clinical Study Report No. CA13895

#### Appendices 16.2.8.2 to 16.2.8.6 will have the following format.

Appendix 16.2.8.1 Clinical Laboratory Report - Serum Chemistry


| Subject<br>Number | Age/<br>Gende: | Study<br>r Period | Treatment | Hour | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) | Parameter6<br>< Range><br>(Unit) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| X | XX | Screen | | | DDMMYYYY | XX HN | XX | XX | XX | XX HN | XX | _ |
| | XX | X | X | | DDMMYYYYY | XX LY | XX LN | XX | XX LY | XX | XX | |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study.

Note: H = Above Reference Range, L = Below Reference Range
Computer: N = Not Clinically Significant, Y = Clinically Significant
PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event
Treatment A = 60 mg WTX101 on Day 1 (Fasted)
Treatment B = 60 mg WTX101 on Day 1 (Fed)
Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895

Appendix 16.2.8.7 Clinical Laboratory Report - Comments


| Subject<br>Number | | Treatment | Hour | Date | Department | Test | Result | Unit | Comment |
|---|---|---|---|---|---|---|---|---|---|
| X | X | X | -X.X I | DD <b>MM</b> MYYYY | Other Tests | Fibrinogen | XXX | mg/dL | Not significant in the |

Note: Treatment A = 60 mg WTX101 on Day 1 (Fasted) Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

## Celerion, Clinical Study Report No. CA13895

Appendix 16.2.9.1 Vital Signs

| D ~- | 1 | ~ f | 7.7 |
|------|-----|-----|-----|
| Page | - 1 | () | X |

| | | | | | | | ] | Blood 1 | Pressure (mmHg) | | Respir- | Temper- | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | | Treatment | Day | Hour | Date | Time | | | Systolic/Diastolic | | ation<br>(rpm) | ature<br>(C) | Weight<br>(kg) | Comments |
| Х | Screen | | • | | DDMMYYYY | X:XX:XX | | | | | | | XXX.X | |
| | | | | | DDMMYYYYY | X:XX:XX | SITX | Right | XXX/ XX | XX | XX | XX.X | | |
| | X | X | -X | -XX.X | DDMMYYYYY | XX:XX:XX | SITX | Right | XXX/ XX | XX | XX | XX.X | | |
| | | | X | -X.X | DDMMYYYYY | X:XX:XX | SITX | Right | XXX/ XX | XX | XX | XX.X | | |
| | | | | X.X | DDMMYYYYY | X:XX:XX | SITX | Right | XXX/ XX | XX | XX | XX.X | | |
| | | | | XX.X | DDMMMYYYY | XX:XX:XX | SITX | Right. | XXX/ XX | XX | XX | XX.X | | |

Note: SITX = X-minute sitting, R = Recheck Value.

Treatment A = 60 mg WTX101 on Day 1 (Fasted)

Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

## Celerion, Clinical Study Report No. CA13895

### Appendix 16.2.9.2 12-Lead Electrocardiogram

| Page | 1 | of | V |
|------|---|----|---|
| raye | | OT | Δ |

| | oject Study<br>Mber Period | Treatment | Day | Hour | Date | Time | Result | Heart<br>Rate<br>(bpm) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTCB*<br>(msec) | QTCF*<br>(msec) Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| X | Screen | | | | DDMMYYYY | X:XX:XX | Normal | XX | XXX.X | XX.X | XXX.X | XXX.X | XXX.X |
| | Y | V | V | Y Y | | V • VV • VV | Abnormal NCS | VV | VVV V | XX X | YYY Y | YYY Y | XXX X |

Note:  $QTcB^* = QTc$  corrected using Bazzet's correction,  $QTcF^* = QTc$  corrected using Fridericia's correction.

NCS = Not clinically significant

Treatment A = 60 mg WTX101 on Day 1 (Fasted) Treatment B = 60 mg WTX101 on Day 1 (Fed)

Treatment C = 20 mg omeprazole QD on the morning of Days -5 to -1 (Fasted), 20 mg omeprazole capsule at Hour -1 and 60 mg WTX101 at Hour 0 on Day 1 (Fasted)

WTX101: WTX101-102

Celerion, Clinical Study Report No. CA13895


Appendix 16.2.9.3 Phone Participant

| Subject | Study | | | | | |
|---|---|---|---|---|---|---|
| Number | Period | Time Point | Date | Time | Result | Comments |
| X | A11 | First attempt | DDMMMYYYY | 'HH:MM | XXXXX | XXXXXXXXXXX |